# 16.1.9 Documentation of Statistical Methods

MRT5005-101 Final Statistical Analysis Plan, Version 1.0, 26 October 2021

NCT Number: NCT03375047

# STATISTICAL ANALYSIS PLAN 26 October 2021 FINAL v1.0

A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled, Combined Single and Multiple Ascending Dose Study Evaluating the Safety, Tolerability, and Biological Activity of MRT5005 ( mRNA LNP) Administered by Nebulization to Adult Subjects with Cystic Fibrosis

PROTOCOL NUMBER MRT5005-101 Version 5.0, Amendment 4

SPONSORED BY

Translate Bio, Inc. 29 Hartwell Avenue Lexington, MA 02421

PREPARED BY

Rho, Inc. 2635 E NC Hwy 54 Durham, NC 27713 Telephone: (919) 408-8000

Fax: (919) 408-0999

This document is confidential and proprietary to **Translate Bio, Inc.** Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein will be reproduced, published, or otherwise disclosed without the prior written approval of **Translate Bio, Inc.**, except that this document may be disclosed to appropriate Institutional Review Boards under the condition that they keep the information confidential.

Statistical Analysis Plan 26 October 2021

# **DOCUMENT VERSION CONTROL**

| Version Number | Date | Comments/Changes |
|----------------|-----------------|------------------|
| 1.0 | 26 October 2021 | Initial Version |

## **APPROVALS**

| _ | |
|-----------|--------------------------------------|
| Approved: | |
| | Vice President, Clinical Development |
| _ | Translate Bio, Inc. |
| | Manager, Clinical Trials |
| | Translate Bio, Inc. |

Principal Biostatistician

Rho, Inc.

# **TABLE OF CONTENTS**

| LIS | T OF ABBREVIATIONS | 6 |
|---|---|---|
| 1. | PURPOSE OF THE ANALYSES | 7 |
| 2. | PROTOCOL SUMMARY | 8 |
| | 2.1 Study Objectives | |
| | 2.1.1 Primary Objective | |
| | 2.1.2 Secondary Objective | |
| | 2.2 Study Endpoints | 8 |
| | 2.2.1 Primary Endpoint | |
| | 2.2.2 Secondary Endpoint | |
| | <ul><li>2.3 Overall Study Design and Plan</li><li>2.4 Treatment Regimens and Randomization</li></ul> | |
| | <ul><li>2.4 Treatment Regimens and Randomization</li><li>2.5 Sample Size Determination</li></ul> | |
| | 2.6 Protocol Safety Review Committee | |
| | 2.7 Dose Group and Study Stopping Criteria and Unblinding | |
| 3. | GENERAL ANALYSIS AND REPORTING CONVENTIONS | |
| | ANALYSIS SETS | |
| 4. | | |
| | 4.1 Safety Analysis Set | |
| <b>5</b> . | STUDY PATIENTS | |
| | 5.1 Disposition of Patients | |
| | 5.2 Protocol Deviations | . 18 |
| <b>6</b> . | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 19 |
| <b>7</b> . | MEASUREMENTS OF TREATMENT COMPLIANCE | 20 |
| 8. | EFFICACY EVALUATION | 21 |
| 9. | SAFETY EVALUATION | . 22 |
| | 9.1 Overview of Safety Analysis Methods | |
| | 9.2 Extent of Exposure | |
| | 9.3 Adverse Events | |
| | 9.3.1 Overall Summary of AEs | 23 |
| | 9.3.2 Subject-level and Event-level Summary of AEs | |
| | 9.4 Deaths, Serious Adverse Events, and Other Significant Adverse Events | |
| | <ul><li>9.5 Clinical Laboratory Evaluation</li></ul> | |
| | 9.6.1 Vital Signs | |
| | 9.6.2 Physical Examinations | |
| | 9.6.3 Other Safety Measures | |
| | 9.6.3.1 Electrocardiogram Findings | 26 |
| | 9.6.3.2 Spirometry | |
| | 9.6.3.3 Chest X-ray | |
| | 9.6.3.4 Prior and Concomitant Medications and Procedures | |
| | 9.6.3.5 Serum Inflammatory Markers | |
| 10. | PHARMACOKINETIC EVALUATION | . 29 |

| 11. | OTHER ANALYSES | 30 |
|-------------|----------------------------------------------------|----|
| | 11.1 Cystic Fibrosis Questionnaire-Revised (CFQ-R) | 30 |
| <b>12</b> . | CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL | 31 |
| 13. | REFERENCES | 32 |
| 14. | LIST OF PLANNED TABLES | 33 |
| <b>15</b> . | LIST OF PLANNED FIGURES | 39 |
| <b>16</b> . | LIST OF PLANNED DATA LISTINGS | 42 |
| <b>17.</b> | APPENDICES | 46 |
| | 17.1 Study Flow Chart | 46 |
| | 17.2 Subject Enrollment and Treatment Allocation | |
| | 17.3 Schedule of Events | |
| 18. | ATTACHMENTS | 49 |

#### LIST OF ABBREVIATIONS

AE adverse event
BMI body mass index
CF cystic fibrosis

CFQ-R cystic fibrosis questionnaire-revised

CFTR cystic fibrosis transmembrane conductance regulator

CSR clinical study report

ECG electrocardiogram

FEF forced expiratory flow

FEV<sub>1</sub> forced expiratory volume in 1 second

hCFTR human cystic fibrosis transmembrane conductance regulator

ICH International Council for Harmonisation

MAD multiple ascending dose

MedDRA Medical Dictionary for Regulatory Activities

PEF peak expiratory flow

PSRC Protocol Safety Review Committee qPCR quantitative polymerase chain reaction

SAD single ascending dose
SAE serious adverse event
SAP statistical analysis plan

SD standard deviation

SUSAR suspected unexpected serious adverse reaction

TEAE treatment-emergent adverse event

ULN upper limit of normal

## 1. PURPOSE OF THE ANALYSES

The statistical analysis plan (SAP) is being developed after review of the Translate Bio, Inc., protocol number MRT5005-101, but before the final analyses of the data. The SAP contains detailed information to aid in the implementation of the statistical analyses and reporting of the study data for use in the clinical study report (CSR).

This SAP is being written with due consideration of the recommendations outlined in the most recent International Council for Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the analysis sets that will be analyzed, the subject characteristics parameters, and the safety parameters that will be evaluated. The details of the specific statistical methods that will be used are provided in the SAP. Table, figure, and listing specifications are provided in separate documents.

## 2. PROTOCOL SUMMARY

# 2.1 Study Objectives

## 2.1.1 Primary Objective

To evaluate the safety and tolerability of single and multiple escalating doses of MRT5005 administered by nebulization to adult subjects with cystic fibrosis (CF).

# 2.1.2 Secondary Objective

To evaluate the effect on percent predicted forced expiratory volume in 1 second (ppFEV<sub>1</sub>) and other spirometry parameters after single and multiple escalating doses of MRT5005 administered by nebulization to adult subjects with CF.

## 2.2 Study Endpoints

## 2.2.1 Primary Endpoint

The safety and tolerability of nebulized MRT5005 will be assessed based on the types, frequency, and severity of treatment-emergent AEs including pulmonary exacerbations; concomitant medication use; and changes from baseline in physical examination, weight, vital signs, oxygen saturation (pulse oximetry), ECG, standard clinical laboratory tests, chest x-ray, and spirometry as a measure of pulmonary function.

# 2.2.2 Secondary Endpoint

The biological activity of nebulized MRT5005 will be assessed based on changes from baseline in ppFEV $_1$  and other spirometry parameters.

# 2.3 Overall Study Design and Plan

This phase 1/2 study is designed as a randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial, which will be conducted in 3 parts. Subjects will be administered single and multiple escalating doses of MRT5005 in Parts A and B of the study, respectively. In Part D, subjects will be administered 5 consecutive daily doses of 4 mg MRT5005 or placebo. Part C (bronchoscopy groups) was removed from the protocol in the 3rd amendment to the protocol (Version 4.0 dated 29 July 2019).

The study will be conducted at multiple centers in the United States with expertise in treating CF subjects. At least 40 adult male and female subjects with CF, 18 years of age or older, are planned to participate in the study. Subjects who are clinically stable with a forced expiratory volume in 1 second (FEV<sub>1</sub>)  $\geq$ 50% and  $\leq$ 90% predicted, and who meet all inclusion criteria and none of the exclusion criteria, will be eligible for the study. The inclusion and exclusion criteria for the study are enumerated in Sections 4.1 and 4.2 of the protocol, respectively. Women of childbearing potential will also be eligible to participate if they are willing and able to comply with contraception requirements.

If subjects do not complete the study or complete certain procedures, additional subjects will be enrolled at the Sponsor's discretion to ensure that at least 16, 16, and 8 evaluable subjects complete Parts A, B, and D of the study, respectively. For Part A, an evaluable subject will be defined as a subject with 1 completed dose and 4 weeks of safety follow-up. For Part B, an evaluable subject will be defined as a subject with 4 completed doses occurring on 4 consecutive weeks with 4 weeks of safety follow-up. For Part D, an evaluable subject will be defined as a subject with 4 completed doses occurring within 5 consecutive days with 4 weeks of safety follow-up. A SAD dose group may be repeated in a new group of subjects in Part A to further assess the safety of the dose level before escalating to the next higher dose level, or before allowing it to proceed from Part A (SAD) to Part B (MAD). It is expected that no more than 1 additional group of 4 subjects will be enrolled into the study in Part A. Therefore, up to a maximum of 44 evaluable subjects may participate in the study.

Each part of the study will consist of a screening period, a treatment period, and a follow-up period. Multiple visits during the screening period, from Day -28 to Day -2 (Parts A and B) or from Day -28 to Day -1 (Part D), may be necessary for the subject to complete all of the required screening procedures and tests. During the treatment period, subjects participating in Part A will be confined to the study center from Day -1 to Day 2 and will receive a single dose of investigational product. This will be followed by a safety follow-up period, which continues up to the final study visit on Day 337. During the safety follow-up, clinic visits for Part A subjects will be performed on an outpatient basis.

No confinement will be required of subjects in Parts B and D of the study; these subjects will perform all clinic visits in the treatment and follow-up periods as outpatients. During the treatment period of Part B (Day -1 to Day 33), subjects will receive 5 doses of investigational product, administered 1 dose per week for 5 weeks. During the treatment period of Part D (Day 1 to Day 5), subjects will receive 5 doses of IP, administered 1 dose per day for 5 days. The safety follow-up period will continue up to the last study visit on Day 365 for Part B and Day 341 for Part D.

In Part A (SAD groups), 4 groups consisting of 4 subjects each will be enrolled sequentially to receive single doses of MRT5005 or placebo (normal saline) administered by nebulization. Three dose levels of MRT5005 were planned to be investigated: 8, 16, and 24 mg of

mRNA (the active drug substance of MRT5005; nominal doses)]. An additional treatment group (20 mg) was added after blinded safety information from the 24 mg dose group revealed the occurrence of febrile reactions in 3 of 4 subjects. Within each dose group, the enrollment and treatment of the 4 subjects will be staggered by at least 1 week. Subjects will be randomized in a 3:1 ratio to receive a single dose of either MRT5005 or placebo (3 subjects to receive MRT5005 and 1 subject to receive placebo per dose group).

The protocol safety review committee (PSRC) will be responsible for reviewing safety data and, based on this review, making the decision to dose escalate from the 8 mg starting SAD dose level to the 16 mg dose level, and then to the 24 mg maximum dose level. The 20 mg dose level will be evaluated after the 24 mg dose level.

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx

mRNA [

Statistical Analysis Plan

26 October 2021

The decision to begin enrollment and treatment of the initial 8 mg multiple-dose group in Part B will also be made by the PSRC, based on a review of at least 28 days of safety follow-up for all subjects who received a single dose of the 8 mg dose level in Part A.

In Part B (MAD groups), 4 groups consisting of 4 subjects each will be enrolled sequentially to receive multiple doses of MRT5005 or placebo administered by nebulization. Three groups will be enrolled sequentially to receive dose levels of MRT5005 investigated as single doses in Part A (8, 16, and 20 mg). An additional dose level that was not investigated in Part A (12 mg) will also be evaluated in Part B. The 12 mg dose group may be enrolled in parallel with the 16 and/or 20 mg dose group. Within each dose group, subjects will be randomized in a 3:1 ratio to receive 5 doses of either MRT5005 or placebo (3 subjects to receive MRT5005 and 1 subject to receive placebo per dose group), administered 1 dose per week for 5 weeks. The enrollment and treatment of the 4 subjects within each dose group will be staggered by at least 2 weeks (the next subject in the dose group will be enrolled and treated only when the previous subject has received their second dose and at least 1 week of safety follow-up), with the exception of the 12 mg dose group in Part B which may not require staggered treatment as outlined in Protocol Section 3.1.

Similar to Part A, the PSRC will be responsible for reviewing safety data and making the decision to dose escalate.

In Part D, 8 subjects will be randomized in a 3:1 ratio to receive 5 doses of either 4 mg MRT5005 or placebo, administered at 1 dose per day for 5 consecutive days.

Because single doses up to 20 mg, as well as 5 weekly doses up to 16 mg have been tolerated in Parts A and B, the enrollment and treatment of the 8 subjects within Part D will not be staggered.

All subjects in the study will be monitored for safety for 12 months after administration of the last dose of investigational product (post-single dose in Part A; post-fifth dose in Parts B and D). The safety and tolerability of nebulized MRT5005 will be assessed based on the types, frequency, and severity of treatment-emergent adverse events (TEAEs) reported including the number of pulmonary exacerbations; concomitant medication use; and changes from baseline in physical examination, weight, vital signs, oxygen saturation (pulse oximetry), electrocardiogram (ECG), standard clinical laboratory tests, chest x-ray, and spirometry as a measure of pulmonary function. As part of the safety evaluation, assays to detect in the blood post-treatment will be performed along with assays to detect antibody and T cell immune responses to CFTR protein and anti-PEG (polyethylene glycol) antibodies.

This will be conducted as a double-blind study, except for the last part of the 12-month follow-up. All subjects in the study will be followed up for 12 months after their last dose, but the treatment randomization for the 8, 16, and 24 mg single dose groups will be unblinded 1 month after the last dose of the last subject in the 24 mg single dose group in Part A. The blind will be maintained in the 20 mg single dose group in Part A, as well as the 8, 16, and 12 mg multiple dose groups in Part B until the 1-month time point after the last dose (Day 57) of

the last subject dosed in the 12 mg dose group. For the 20 mg multiple dose group in Part B, the blind will be maintained until the last subject in this group has reached the 1-month time point after the last dose day (Day 57). For Part D, the blind will be maintained until the 1month time point after the last dose (Day 32) of the last subject in Part D.

During the double-blind period, the investigators and all study staff involved in the evaluation of subject eligibility, administration of IP, and assessment of the study outcomes will be blinded to treatment assignment (MRT5005 vs. placebo within each dose group) until planned unblinding. All subjects and their families, as well as sponsor personnel in direct contact with the study center, will also be blinded.

A study flow chart is presented in Appendix 17.1, and a flow diagram of subject enrollment and treatment allocation is presented in Appendix 17.2. Table 1 through Table 9 in the protocol present the schedule of study procedures to be performed during each the 3 periods in Part A, B, and D of the study.

## **Treatment Regimens and Randomization**

In all three parts of the study, subjects will be randomized to receive either MRT5005 or placebo (normal saline) in a 3:1 ratio. Subjects will receive a single dose in Part A, 5 weekly doses in Part B, and 5 consecutive daily doses in Part D. The 8 mg dose level of MRT5005 will be the SAD starting dose in Part A followed by sequential escalation to the 16 mg and 24 mg dose levels of MRT5005. An additional 20 mg treatment group was added to Part A after blinded safety information from the 24 mg group revealed the occurrence of febrile reactions in 3 of 4 subjects. The 8 mg dose level of MRT5005 will be the MAD starting dose in Part B, followed by sequential escalation to the 16 mg and 20 mg dose levels of MRT5005. An additional 12 mg group was added to Part B to explore the safety profile at an intermediate dose level that was not investigated as a single dose in Part A. The 12 mg dose level may begin enrollment in parallel with the 16 mg dose level. The enrollment and treatment of the 4 subjects within each MAD dose group will be staggered by at least 2 weeks (the next subject in the dose group will only be enrolled and treated when the previous subject has received their second dose and there is approximately 1 week of safety follow-up), with the exception of the 12 mg dose group in Part B which may not require staggered treatment. In Part D, 8 subjects will be randomized in a 3:1 ratio to receive 5 doses of either 4 mg MRT5005 or placebo, administered at 1 dose per day for 5 consecutive days. Because single doses up to 20 mg, as well as 5 weekly doses up to 16 mg have been tolerated in Parts A and B, the enrollment and treatment of the 8 subjects within Part D will not be staggered. During the treatment of subjects in Part D, should AEs occur that indicate the study drug is not tolerated well, the enrollment and treatment of subjects may be terminated by the PSRC and Sponsor, and enrollment and treatment of a lower dose strength may be considered in the remaining subjects in the cohort. For example, if the tolerability of the 4 mg daily dose level is found to be unacceptable, then the 2 mg dose level can be considered for investigation. Subjects will not be allowed to participate in more than 1 part of the study.

## 2.5 Sample Size Determination

The sample size is not based on any statistical considerations. Instead, the sample size is based on traditional phase 1 first-in-human study designs for this disease population. In Parts A and B of the study, the inclusion of 4 subjects per dose group (3 subjects randomized to MRT5005 and 1 subject randomized to placebo) will provide basic information on safety and tolerability during dose escalation of MRT5005. In Part D, 8 subjects treated at 4 mg MRT5005 or placebo (6 subjects randomized to MRT5005 and 2 subjects randomized to placebo) will provide further safety and tolerability data on MRT5005. This study is also designed with the flexibility to enroll additional groups of subjects to support meeting its objectives.

# 2.6 Protocol Safety Review Committee

The PSRC will conduct a safety data review before each dose-escalation in Parts A and B and before the initiation of enrollment and treatment of subjects in the first MAD group in Part B. Based on these safety data reviews, the PSRC will decide whether or not to proceed at each of these time points in the study, per Protocol Sections 3.4.1 and 3.4.2.

Based on the judgment of the PSRC:

• A Part A dose group may be repeated in a new group of subjects to further assess the safety of the dose level before escalating to the next higher dose level or before multiple dosing is allowed to proceed in Part B.

The PSRC will be notified of all serious adverse events deemed possibly, probably, or definitely related to investigational product (including suspected unexpected serious adverse reaction [SUSAR]) reports in real-time. The PSRC will be notified of 2 occurrences of significant febrile reactions in different participants (defined as ≥ Grade 2 fever [>39.0°C] associated with systemic symptomatology [eg, body aches, malaise, nausea]) within 24 hours following administration of IP. If an adverse event of special interest (AESI), as defined in Protocol Section 8.1.8, is reported during the study, the PSRC will be notified by the Sponsor in real-time. The PSRC will receive SAE listings following each dose group and may choose to receive more frequent SAEs listings at any time during the study. The PSRC will also review all available and relevant safety data if stopping criteria are met during the study to determine whether the study will continue or be terminated. The PSRC charter includes the roles and responsibilities of the PSRC, format and structure of PSRC meetings, and details the study stopping criteria.

## 2.7 Dose Group and Study Stopping Criteria and Unblinding

Investigational product administration will be halted for all subjects in a dose group, as well as any subjects in an ongoing higher dose group if any of the following stopping criteria are met:

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 

#### CONFIDENTIAL

- a. Two subjects in a dose group experience a significant febrile reaction (defined as ≥ Grade 2 fever [>39.0°C] associated with systemic symptomatology [eg, body aches, malaise, nausea]) within 24 hours following administration of IP.
- b. Two subjects in a dose group experience a suspected moderate to severe allergic/hypersensitivity reaction, including but not limited to anaphylaxis, generalized rash, edema or bronchospasm possibly related to drug treatment.

Investigational product administration will be halted for all subjects in Part D if the following stopping criterion is met:

a. Three subjects experience Grade 1 fevers (38.0 to 39.0 °C) associated with systemic symptomatology (eg, body aches, malaise, nausea) onset within 24 hours following administration of IP on ≥3 separate occasions.

Investigational product administration will be halted for all subjects if any of the following stopping criteria are met:

- a. A subject experiences a Grade 4, life-threatening treatment-emergent AE or death that is considered probably or definitely related to investigational product by the Investigator.
- b. Two or more subjects in a dose group experience 1 or more moderate or severe pulmonary exacerbations during the 5-week treatment period in part B or through Day 11 (1 week post-5<sup>th</sup> dose) in Part D.
- c. Two or more subjects in a dose group experience a decrease in predicted FEV1 of at least 25 % compared to the baseline value (defined as the average of the Day -1 and Day 1 pre-dose values) during the 5-week treatment period in Part B or through Day 11 (1 week post-5<sup>th</sup> dose) in Part D that cannot be explained, in the opinion of the PI, by the underlying disease of CF and that is confirmed on 2 separate occasions at least 3 days apart.
- d. Two or more subjects in the study experience a suspected serious allergic/hypersensitivity reaction, including but not limited to anaphylaxis, generalized rash or bronchospasm likely to be related to drug treatment.
- e. Two or more subjects in a dose group experience a deterioration in liver function, as detailed below:
  - i. Elevation of ALT or AST to >5x ULN in a subject regardless of baseline value
  - ii. Elevation of ALT or AST to >3x ULN in a subject with a normal baseline or elevation of >3x ULN from the subject's actual baseline if not normal, with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).
  - iii. Elevation of ALT or AST to >3x ULN in a subject with a normal baseline or elevation of >3x ULN from the subject's actual baseline if not normal, and total bilirubin >2x ULN or INR >1.5.

To determine whether these stopping rules have been met, the relevant data will be reviewed by the PSRC. To ensure subject safety, the PSRC may request unblinding the treatment assignment(s) for an individual subject or for an entire dose group.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 


#### 3. GENERAL ANALYSIS AND REPORTING CONVENTIONS

The following is a list of general analysis and reporting conventions to be applied for this study. Where appropriate, clarification is provided throughout this SAP to document planned differences for analyses by study part.

Categorical variables will be summarized using counts (n) and percentages (%) and will be presented in the form "n (xx.x)." If a count is 0, 0% will be shown for the percentage. To ensure completeness, summaries for categorical and discrete variables will include all categories, even if no subjects had a response in a particular category.

Continuous variables will be summarized using number of subjects (n), value for each subject, mean, and SD. The mean will be reported to 1 more level of precision than the original observations, and the SD will be reported to 2 more levels of precision than the original observations, up to a maximum of 4 decimal places.

All analyses will be performed using SAS® System version 9.4 or later.

Dates in listings will be displayed as yyyy-mm-dd (e.g., 2015-01-24).

In general, age will be calculated in years using the date of birth and the date of informed consent as [(date of informed consent – date of birth)]/365.25, rounded down to the next largest integer using the floor function.

Unless otherwise specified, the baseline value for all measures is the last non-missing value prior to the first dose, obtained on or before the date of the first dose of study drug. For measurements that occur on the date of the first dose of study drug with time collected, the measurement will be considered the baseline value if the measurement time is prior to the time of the first dose. The average of the results from the testing on Day -1 and at pre-dose on Day 1 will serve as the subject's baseline for spirometry testing for Part A and Part B. For Part D, the Day 1 pre-dose result will serve as the subject's baseline ECG for Part A and Part B. For Part D, the screening ECG will serve as the subject's baseline ECG.

For any laboratory values containing an inequality in the result, the numeric portion of the result will be used for analysis (e.g., <0.1 will be treated as 0.1).

Unless otherwise specified, each display will be presented separately for each study part. For any by study part displays categorized by dose group, summaries will show columns for the 4 mg dose group, 8 mg dose group, 12 mg dose group, 16 mg dose group, 20 mg dose group, 24 mg dose group, and a pooled placebo group, as applicable for each study part. A total column will be displayed where applicable.

Where possible and when specified, integrated displays will be presented combining data from all study parts by treatment (all active MRT5005 treatment dose groups combined, all pooled placebo groups combined).

For any by study part displays categorized by dose group, summaries will show columns for the 4 mg dose group, 8 mg dose group, 12 mg dose group, 16 mg dose group, 20 mg dose group, 24 mg dose group, and a pooled placebo group, as applicable for each study part. A total column will be displayed where applicable.

All data listings and figures will be presented by study part, unless otherwise specified.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 

## 4. ANALYSIS SETS

# 4.1 Safety Analysis Set

The primary analysis population for safety will be the safety analysis set, which will include all randomized subjects who received investigational product. For all safety analyses, subjects will be analyzed according to the treatment they actually received.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 

#### 5. STUDY PATIENTS

## 5.1 Disposition of Patients

The disposition of subjects will be summarized for all subjects screened in the study. The following disposition information will be summarized overall for each study part, and for the study overall:

• The number and percentage of subjects that were screened, randomized, that were screen failures, and the reason for screen failure

The following disposition information will be summarized for the safety analysis set for each study part by dose group, and for the study overall by pooled treatment group:

- The number and percentage of subjects who completed the study
- The number and percentage of subjects who discontinued the study and the reason for premature discontinuation

A data listing of subject disposition for all subjects in the safety analysis set and a data listing of screen failures for all screened subjects will also be provided.

A data listing of visits not done, or completed as a home health visit or telephone visit as a replacement for a scheduled in-clinic visit and the corresponding reason for all subjects in the safety analysis set will be provided.

#### 5.2 Protocol Deviations

Protocol deviations for all subjects in the safety analysis set will be summarized for each study part by type and dose group. A data listing of all protocol deviations for all subjects in the safety analysis set will also be provided.

#### 6. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Subject demographics and other baseline characteristics will be summarized descriptively for the safety analysis set for each study part, and for the study overall by pooled treatment group. The demographic and baseline characteristic summaries will be used to describe the study population.

Demographic data will include age, sex, race, ethnicity, baseline percent predicted  $FEV_1$ , concomitant CFTR modulator use, and genotype. Genotype will be summarized by first mutation class and second mutation class (e.g., 'Class I/Class II'). Age (years) will be calculated using the date of birth and the date of informed consent, as described in Section 3.

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 23.1 to identify the system organ class and preferred term. A summary table will be presented by dose group to reflect a count of medical history events occurring in subjects in the safety analysis set within each system organ class and preferred term for each study part, and for the study overall. All percentages will use the number of subjects in the safety analysis set as the denominator. Therefore, if a subject has more than 1 medical history event within a system organ class, the subject will be counted only once in that system organ class. If a subject has more than 1 medical history event that codes to the same preferred term, the subject will be counted only once for that preferred term. Tabular summaries will be sorted by overall (MRT5005 + Placebo) descending frequency by system organ class and by preferred term.

Individual data for demographics and medical history will be presented in the data listings for subjects in the safety analysis set.

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 

## 7. MEASUREMENTS OF TREATMENT COMPLIANCE

Treatment compliance and exposure to investigational product will be summarized in terms of number of doses (total, full, and partial) administered. The number and percentage of subjects with 1, 2, 3, 4, or 5 total doses (sum of full and partial) administered will be presented by dose group for each study part, and by pooled treatment group for the study overall. The number of full doses and partial doses administered will be separately summarized continuously using descriptive statistics by dose group for each study part, and by pooled treatment group for the study overall. The number of full doses administered is the number of individual occurrences (days) for which a subject received a full dose of investigational product based on the completion of nebulization for the expected number of medication chambers, even if there was excess residual observed in the chamber after completion of nebulization. A partial dose refers to incomplete nebulization. Full and partial doses are independent of the presence or absence of excess residual in the medication chamber.

Individual data for dosing, including the start and end dates and time of nebulization along with assessments of whether nebulization was complete and whether excess residual was present in the medication chamber will be listed by visit and nebulizer for subjects in the safety analysis set. The number of full doses and partial doses administered for each subject will be presented in a data listing for subjects in the safety analysis set. The following individual data for dosing for each subject at each visit will be presented in a data listing for subjects in the safety analysis set: date of IP administration, whether full dose was administered, reason if full dose not administered, actual number of medication chambers completed, and the expected number of medication chambers completed.

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 

# 8. EFFICACY EVALUATION

Not applicable.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 

#### CONFIDENTIAL

#### 9. SAFETY EVALUATION

## 9.1 Overview of Safety Analysis Methods

The safety analyses will be performed using the safety analysis set for the safety measures, which include extent of drug exposure, adverse events (AEs), vital signs, clinical laboratory data, ECGs, pulse oximetry, chest x-rays, spirometry, physical examinations, concomitant medications, and serum inflammatory markers.

Safety data will not be imputed, except for partial dates, which will be imputed only for defining TEAEs and for the calculation of the duration of the AE. Completely missing dates will not be imputed and any AE with a completely missing date will be classified as a TEAE. Imputed dates will not be presented in data listings.

Partial dates will be imputed for the purposes of defining TEAEs as follows:

- For a missing start day where the month and year are present, the start day will be set to the first day of the month, unless 1) the first day of the month is before the date of first dose of study drug and the month and year are the same as the month and year of the date of first dose of study drug, and 2) the end date is on or after the date of first dose of study drug or the end date is completely missing, in which case the start day will be set to the first day of first dose of study drug.
- For a missing start day and month where the year is present, the start day and month will be set to January 1<sup>st</sup>, unless 1) January 1<sup>st</sup> is before the date of first dose of study drug and the year is the same as the year of the date of first dose of study drug, and 2) the end date is on or after the date of first dose of study drug or the end date is completely missing, in which case the start day and month will be set to that of the date of first dose of study drug.
- For a missing end day where the month and year are present, the end day will be set to the last day of the month, unless the month and year are the same as the month and year of the last contact date for the subject, in which case the end day will be set to that of the subject's last contact date.
- For a missing end day and month where the year is present, the end day and month will be set to the subject's last contact date, unless the year of the subject's last contact date is greater than the end year, in which case the end day and month will be set to December 31st.

## 9.2 Extent of Exposure

Extent of exposure and treatment compliance are described in Section 7.

#### 9.3 Adverse Events

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 23.1 to identify the system organ class and preferred term.

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 

Treatment-emergent AEs are defined as events that are newly reported or reported to worsen in severity after the start of treatment. Adverse events that occur after the treatment start date, occur on the treatment start date with a time that is equal to or after treatment start time, or that have a missing AE start date will be categorized as treatment-emergent. Treatment-emergent AEs will be summarized for the safety analysis set.

For summaries of TEAEs by time interval, the categorizations for Part A will be: Overall, Study Day 1,  $1 < \text{Study Day} \le 7$ ,  $1 \le \text{Study Day} \le 29$ , and Study Day > 29. The categorizations for Part B will be: Overall, Study Day 1,  $1 < \text{Study Day} \le 7$ ,  $1 \le \text{Study Day} \le 36$ ,  $1 \le \text{Study Day} \le 57$ , and Study Day > 57. The categorizations for Part D will be: Overall, Study Day 1,  $1 < \text{Study Day} \le 5$ ,  $1 \le \text{Study Day} \le 11$ ,  $1 \le \text{Study Day} \le 32$ , and Study Day > 32. The categorizations for the study overall will be: Overall, through 1 month post-dose (Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively), after 1 month post-dose (> Day 29, > Day 57, and > Day 32 for Part A, Part B, and Part D, respectively). Any TEAE with a completely missing start date will not be categorized into a specific time interval, but will be included in the Overall category.

Any dose limiting toxicities identified will be addressed in the clinical study report (CSR).

## 9.3.1 Overall Summary of AEs

An overall summary of AEs will be presented by dose group and will reflect a count of TEAEs, treatment-emergent serious adverse events (SAEs), TEAEs by relationship to investigational product, and TEAEs by severity. Additionally, the table will reflect the count and percentage of subjects experiencing the following: any TEAEs, SAEs, TEAEs leading to treatment discontinuation, TEAEs resulting in death, TEAEs classified as pulmonary exacerbations (investigator and protocol-defined), TEAEs classified by relationship to investigational product, TEAEs classified by relationship to nebulization/treatment administration, and TEAEs by severity. The overall summary of AEs will be presented for the overall time period for each study part, as well as for the study overall. The overall summary of AEs will also be presented for the overall time period and through 1 month post-dose (Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively) by pooled treatment group. All percentages will use the number of subjects in the safety analysis set as the denominator.

# 9.3.2 Subject-level and Event-level Summary of AEs

A summary table will be presented for each study part by dose group to reflect a count and percentage of subjects experiencing at least 1 TEAE in each system organ class and preferred term and a count of TEAEs occurring in subjects in the safety analysis set within each system organ class and preferred term. All percentages will use the number of subjects in the safety analysis set as the denominator. Therefore, if a subject has more than 1 AE within a system organ class, the subject will be counted only once in that system organ class. If a subject has more than 1 AE that codes to the same preferred term, the subject will be counted only once for that preferred term. For the event-level summaries, subjects experiencing more than 1 AE within a system organ class or preferred term will be counted more than once for that system

organ class or preferred term. Tabular summaries will be sorted by descending overall (MRT5005 + Placebo) frequency in subject counts by system organ class and by preferred term.

Using the same subject-level and event-level counting rules, a summary table of TEAEs by preferred term will be presented for the overall time period by dose group for each study part, as well as separately through Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively. In addition, the summary of AEs by preferred term will be presented for the study overall for the overall time interval and through 1 month post-dose (Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively) by pooled treatment group.

All AEs will be presented in data listings for subjects in the safety analysis set, including a flag to distinguish if the AE was treatment-emergent.

# 9.4 Deaths, Serious Adverse Events, and Other Significant Adverse Events

Treatment-emergent SAEs and adverse events of special interest will be summarized for all subjects in the safety analysis set for each study part by dose group and time interval. Summary tables will be presented by dose group to reflect a count and percentage of subjects experiencing at least 1 TEAE in each system organ class and preferred term (subject-level analysis) and a count of TEAEs (event-level analysis) occurring in subjects in the safety analysis set within each system organ class and preferred term within each AE subset (serious, AESIs). All percentages will use the number of subjects in the safety analysis set as the denominator. Therefore, for the subject-level analysis, if a subject has one or more AE within a system organ class, the subject will be counted only once in that system organ class. If a subject has one or more AE that codes to the same preferred term, the subject will be counted only once for that preferred term. For the event-level analysis, subjects experiencing more than 1 AE within a system organ class or preferred term will be counted according to the number of AEs they experience (more than once) for that system organ class or preferred term. Tabular summaries will be sorted by descending overall (MRT5005 + Placebo) frequency in subject counts by system organ class and by preferred term.

Using the same subject-level and event-level counting rules, treatment-emergent pulmonary exacerbations (investigator and protocol-defined) will be summarized by preferred term for all subjects in the safety analysis set for each study part by dose group and time interval.

Treatment-emergent febrile reactions and hypersensitivity reactions will be presented as a count of febrile reactions, febrile reactions by severity, hypersensitivity reactions, and hypersensitivity reactions by severity. Additionally, the table will reflect the count and percentage of subjects experiencing the following: any febrile reaction, any febrile reaction by severity, any hypersensitivity reaction, and any hypersensitivity reaction by severity. The summary will be for all subjects in the safety analysis set by dose group for each study part. In addition, the summary of treatment-emergent febrile reactions and hypersensitivity reactions will be presented for all subjects in the safety analysis set for the study overall by pooled treatment group. Febrile reactions will be identified based on a preferred term of body temperature increased or preferred term of pyrexia within the 24 hours after completion of

nebulization on any dosing day with at least one other systemic symptom reported as a preferred term of headache, arthralgia, myalgia, fatigue, chills, nausea, or vomiting within the 24 hours after completion of nebulization on any dosing day. Severity grade for febrile reactions will be based on the maximum severity of the preferred terms comprising the febrile reaction. Hypersensitivity reactions will be identified based on a preferred term of hypersensitivity within the 24 hours after completion of nebulization on any dosing day.

Adverse events leading to withdrawal from treatment, AEs resulting in death, pulmonary exacerbations (investigator and protocol-defined), adverse events of special interest, and SAEs will be presented in data listings for subjects in the safety analysis set. Adverse events of pyrexia or body temperature increased during nebulization or within the 24 hours after completion of nebulization on any dosing day will also be listed for subjects in the safety analysis set. This listing will include all adverse events that occurred during nebulization or within the 24 hours after completion of nebulization for subjects that had an adverse event of pyrexia or body temperature increased during nebulization or within the 24 hours after completion of nebulization on any dosing day. All adverse events that occurred during nebulization or within the 24 hours after completion of nebulization will also be listed for subjects in the safety analysis set. Febrile reactions and hypersensitivity reactions within the 24 hours after completion of nebulization on any dosing day will also be listed for subjects in the safety analysis set. This listing will include all adverse events that meet the specified febrile reaction or hypersensitivity criteria that occurred within the 24 hours after completion of nebulization for subjects that had a febrile reaction or hypersensitivity reaction within the 24 hours after completion of nebulization on any dosing day.

# 9.5 Clinical Laboratory Evaluation

Baseline and all post-baseline visit values and change from baseline to post-baseline in laboratory parameters for clinical chemistry and hematology will be summarized for the safety analysis set for each study part by dose group using descriptive statistics, as described in Section 3.

C reactive protein (mg/L), white blood cell (x10^9/L), and neutrophil (%) results for each subject at each visit by dose group for each study part will be provided in a line plot. An additional line plot of C reactive protein (mg/L) results for each subject at each visit by dose group will be provided for visits through Day 29 for Part A, Day 36 for Part B, and through Day 11 for Part D. Time will be represented proportionally on the x-axis.

Hematology, clinical chemistry, urinalysis, and coagulation (Part B and D) laboratory results will be presented in data listings for subjects in the safety analysis set. The listing will include the classification of low, normal, or high, the reference range, and the clinical significance. Classification of low, normal, and high laboratory values in the data listings will be based on the global laboratory reference ranges used across all sites. Clinical significance will be assessed for out of range values based on local laboratory reference ranges. Reference ranges provided in the data listings will be the global laboratory reference ranges used across all sites.

Statistical Analysis Plan 26 October 2021

Pregnancy results will also be presented in a data listing for subjects in the safety analysis set.

# 9.6 Vital Signs, Physical Findings, and Other Observations Related to Safety

## 9.6.1 Vital Signs

Baseline and all post-baseline visit values and change from baseline to post-baseline values in systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, temperature, weight, and pulse oximetry will be summarized for the safety analysis set for each study part by dose group using descriptive statistics, as described in Section 3. Height and body mass index (BMI) at baseline will be summarized for the safety analysis set for each study part by dose group using descriptive statistics, as described in Section 3.

Temperature results for each subject at each visit, through Day 7 for Part A subjects, through Day 36 for Part B subjects, and through Day 11 for Part D subjects, by study part and dose group will be provided in a line plot.

Vital sign results will be presented in a data listing for subjects in the safety analysis set.

## 9.6.2 Physical Examinations

The number and percentage of subjects at each visit with normal, abnormal not clinically significant and abnormal clinically significant physical exam findings for each body system will be summarized for each study part by dose group for the safety analysis set.

Physical examination results will be presented in a data listing for subjects in the safety analysis set.

## 9.6.3 Other Safety Measures

### 9.6.3.1 Electrocardiogram Findings

Shifts from baseline to post-baseline visits for each study part by dose group will be presented for normal, abnormal not clinically significant and abnormal clinically significant ECG findings, as determined by investigator interpretation, for the safety analysis set. Baseline for ECG findings is defined in Section 3.

Electrocardiogram findings will be presented in a data listing for subjects in the safety analysis set.

# 9.6.3.2 Spirometry

Baseline and all post-baseline visit values and change (absolute and relative) from baseline to post-baseline values for FEV<sub>1</sub>, percent predicted FEV<sub>1</sub>, FVC, percent predicted FVC, FEV<sub>1</sub>/FVC, FEF<sub>25-75%</sub>, and PEF will be summarized for the safety analysis set using

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 


descriptive statistics, as described in Section 3. . Baseline for all spirometry parameters is defined in Section 3.

Percent predicted FEV<sub>1</sub> results for each subject at each visit by study part and dose group will be provided in line plots for all visits and separately for visits up to Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively. These plots will be provided by dose group (4) mg [Part D only], 8 mg, 12 mg [Part B only], 16 mg, 20 mg, 24 mg [Part A only], and pooled placebo). Additionally, the mean values with standard error for each of the 4 mg dose group (Part D only), 8 mg dose group, 12 mg dose group (Part B only), 16 mg dose group, 20 mg dose group, 24 mg dose group (Part A only), and pooled placebo group will be provided in a line plot for percent predicted FEV<sub>1</sub> results for all visits and separately for visits up to Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively. The mean change (absolute and relative) from baseline values with standard error for each of the 4 mg dose group (Part D only), 8 mg dose group, 12 mg dose group (Part B only), 16 mg dose group, 20 mg dose group, 24 mg dose group (Part A only), and pooled placebo group will be provided in a line plot for percent predicted FEV<sub>1</sub> results for all post-baseline visits. These line plots will be provided separately for visits up to Day 29, Day 57, and Day 32 for Part A, Part B, and Part D, respectively. Time will be represented proportionally on the x-axis for the Part A and D FEV<sub>1</sub> figures.

Spirometry results will be presented in a data listing for subjects in the safety analysis set.

# 9.6.3.3 Chest X-ray

Shifts from baseline to post-baseline visits for each study part by dose group will be presented for normal, abnormal not clinically significant and abnormal clinically significant assessments for the safety analysis set. Chest x-ray findings will be presented in a data listing for subjects in the safety analysis set.

## 9.6.3.4 Prior and Concomitant Medications and Procedures

The prior and concomitant medications will be coded using the latest version of World Health Organization Drug Dictionary (WHO Drug) Global (2020-SEP) to identify the drug class and preferred drug name.

Concomitant medications will include all medications that started on or after day of first dose of the study drug or that stopped on or after day of first dose of study drug, including medications that are classified as ongoing. Prior medications will include all medications that started and stopped prior to the day of first dose of the study drug. Any medication with a missing stop date (i.e., day, month, and year are missing) will be classified as ongoing. For a medication with a missing start date, the medication will be classified as both a prior and concomitant medication unless the stop date is prior the date of first dose of study drug, in which case the medication will be classified as a prior medication. For medications with start date prior to the date of first dose of study drug and missing end date, the medication will be classified as both prior and concomitant. Medications with missing start and stop dates will be classified as prior and concomitant.

The number and percentage of subjects using prior medications, and separately concomitant medications, will be tabulated by Anatomical Therapeutic Chemical (ATC) level 1 term, ATC level 2 term, and preferred drug name for all subjects in the safety analysis set by study part and dose group, and also for the study overall. If a subject has more than 1 medication within an ATC level 1 term, the subject will be counted only once in that ATC level 1 term. Similarly, if a subject has more than 1 medication within an ATC level 2 term, the subject will be counted only once in that ATC level 2 term. If a subject has more than 1 medication that codes to the same preferred drug name, the subject will be counted only once for that preferred drug name. All percentages will use the number of subjects in the safety analysis set as the denominator. The tabular summaries will be sorted by overall (MRT5005 + Placebo) descending frequency by ATC level 1 term, ATC level 2 term, and preferred drug name.

Prior and concomitant medication data will also be presented in a data listing for subjects in the safety analysis set.

Concomitant surgical procedures will also be presented in a data listing for subjects in the safety analysis set.

# 9.6.3.5 Serum Inflammatory Markers

Serum samples will be analyzed for various inflammatory markers for only Part B 20 mg and Part D subjects.

Baseline and all post-baseline visit values and change from baseline to post-baseline for the inflammatory marker parameters will be summarized for the safety analysis set for each study part by dose group using descriptive statistics, as described in Section 3.

Serum inflammatory marker results will be presented in a data listing for Part B 20 mg and Part D subjects in the safety analysis set.

# **10.PHARMACOKINETIC EVALUATION**

Analyses of pharmacokinetic samples (CFTR mRNA and ) are outside the scope of the SAP.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 

## 11.OTHER ANALYSES

# 11.1 Cystic Fibrosis Questionnaire-Revised (CFQ-R)

For Part B, the CFQ-R respiratory domain scores at baseline (Day -1) and Days 36, 43, 57, 85, 113, 197, 281, and 365 will be summarized for the safety analysis set by dose group using descriptive statistics, as described in Section 3. Change from baseline to post-baseline in CFQ-R respiratory domain scores will be calculated for each subject with data at baseline and the post-baseline visit. The mean change from baseline will be summarized for the safety analysis set by dose group at Days 36, 43, 57, 85, 113, 281, and 365.

CFQ-R respiratory domain scores at each visit will be presented in a data listing for Part B subjects in the safety analysis set.

# 12. CHANGES TO THE ANALYSES PLANNED IN THE PROTOCOL

Not applicable.

Version: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.docx 

## 13. REFERENCES

US Federal Register. (1998) International Conference on Harmonization; Guidance for Industry: Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration. Federal Register, Vol. 63, No. 179, September 16, 1998, page 49583.

US Federal Register. (1996) International Conference on Harmonization; Guidance for Industry: Structure and Content of Clinical Study Reports. Department of Health and Human Services: Food and Drug Administration. Federal Register Vol. 61, July 17, 1996, page 37320.

Version: MRT5005-101 CSR SAP v1.0 26OCT2021.docx 

# **14.LIST OF PLANNED TABLES**

| Rho Table Identifier <sup>a</sup> | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| DM_TAA_F_X | 14.1.1.1 | Summary of Demographic and Baseline Characteristics by Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| DS_TAA_F_X | 14.1.3.1 | Summary of Screen Failures | Screened<br>Subjects | A, B,<br>D, O |
| DS_TAB_F_X | 14.1.3.2 | Summary of Subject Disposition by Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| EX_TAA_F_X | 14.1.4 | Summary of Investigational Product Administration by Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| MH_TAA_F_X | 14.1.5 | Medical History<br>by System Organ<br>Class and<br>Preferred Term by<br>Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| PD_TAA_F_X | 14.1.6 | Protocol Deviations by Type and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAA_F_X | 14.3.1.1 | Overall Summary<br>of Treatment-<br>Emergent Adverse<br>Events by Dose<br>Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAI_F_A | 14.3.1.1.1 | Overall Summary<br>of Treatment-<br>Emergent Adverse<br>Events by Dose<br>Group Through<br>Day 29 | Safety<br>Analysis Set | A |
| AE_TAI_F_B | 14.3.1.1.1 | Overall Summary<br>of Treatment-<br>Emergent Adverse | Safety<br>Analysis Set | В |

| Rho Table Identifier <sup>a</sup> | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| | | Events by Dose<br>Group Through<br>Day 57 | | |
| AE_TAI_F_D | 14.3.1.1.1 | Overall Summary<br>of Treatment-<br>Emergent Adverse<br>Events by Dose<br>Group Through<br>Day 32 | Safety<br>Analysis Set | D |
| AE_TAK_F_O | 14.3.1.1.2 | Overall Summary<br>of Treatment-<br>Emergent Adverse<br>Events by Time<br>Interval | Safety<br>Analysis Set | O |
| AE_TAB_F_X | 14.3.1.2 | Summary of Treatment- Emergent Adverse Events by System Organ Class and Preferred Term by Time Interval and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAC_F_X | 14.3.2.1 | Summary of Treatment- Emergent Serious Adverse Events by System Organ Class and Preferred Term by Time Interval and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAL_F_X | 14.3.2.2 | Summary of Treatment- Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term by Time Interval and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAE_F_X | 14.3.2.3 | Summary of Treatment- | Safety<br>Analysis Set | A, B,<br>D |

| Rho Table Identifiera | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| | | Emergent Adverse Events Classified as Pulmonary Exacerbations by System Organ Class and Preferred Term by Time Interval and Dose Group | | |
| AE_TAH_F_X | 14.3.1.3 | Number of<br>Treatment-<br>Emergent Adverse<br>Events by<br>Preferred Term by<br>Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAJ_F_A | 14.3.1.3.1 | Number of<br>Treatment-<br>Emergent Adverse<br>Events by<br>Preferred Term by<br>Dose Group<br>Through Day 29 | Safety<br>Analysis Set | A |
| AE_TAJ_F_B | 14.3.1.3.1 | Number of<br>Treatment-<br>Emergent Adverse<br>Events by<br>Preferred Term by<br>Dose Group<br>Through Day 57 | Safety<br>Analysis Set | В |
| AE_TAJ_F_D | 14.3.1.3.1 | Number of<br>Treatment-<br>Emergent Adverse<br>Events by<br>Preferred Term by<br>Dose Group<br>Through Day 32 | Safety<br>Analysis Set | D |
| AE_TAN_F_O | 14.3.1.4 | Number of<br>Treatment-<br>Emergent Adverse<br>Events by<br>Preferred Term<br>and Time Interval | Safety<br>Analysis Set | O |
| Rho Table Identifier <sup>a</sup> | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| AE_TAM_F_X | 14.3.2.4 | Summary of Treatment- Emergent Febrile Reactions in First 24 Hours After Completion of Nebulization by Preferred Term and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAO_F_O | 14.3.2.5 | Summary of Treatment- Emergent Febrile Reactions in First 24 Hours After Completion of Nebulization by Preferred Term | Safety<br>Analysis Set | O |
| AE_TAP_F_X | 14.3.2.6 | Summary of Treatment- Emergent Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Preferred Term and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| AE_TAQ_F_O | 14.3.2.7 | Summary of Treatment- Emergent Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Preferred Term | Safety<br>Analysis Set | O |
| LB_TAA_F_X | 14.3.4.1 | Mean and Mean<br>Change from<br>Baseline in<br>Chemistry<br>Laboratory Values | Safety<br>Analysis Set | A, B,<br>D |

| Rho Table Identifier <sup>a</sup> | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| | | by Visit and Dose<br>Group | | |
| LB_TAB_F_X | 14.3.4.2 | Mean and Mean<br>Change from<br>Baseline in<br>Hematology<br>Laboratory Values<br>by Visit and Dose<br>Group | Safety<br>Analysis Set | A, B,<br>D |
| LB_TAE_F_B<br>LB_TAE_F_D | 14.3.4.3 | Mean and Mean<br>Change from<br>Baseline in Serum<br>Inflammatory<br>Markers by Visit<br>and Dose Group | Safety<br>Analysis Set | B, D |
| VS_TAA_F_X | 14.3.5.1 | Mean and Mean<br>Change from<br>Baseline in Vital<br>Signs by Visit and<br>Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| EG_TAA_F_ X | 14.3.6.1 | Shift in Electrocardiogram Findings by Visit and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| CX_TAA_F_X | 14.3.7.1 | Shift in Chest X-<br>Ray by Visit and<br>Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| PE_TAA_F_X | 14.3.8.1 | Summary of Physical Examination by Visit and Dose Group | Safety<br>Analysis Set | A, B,<br>D |
| RE_TAA_F_X | 14.3.9.1 | Mean and Mean<br>Absolute Change<br>from Baseline in<br>Spirometry Values<br>by Visit and Dose<br>Group | Safety<br>Analysis Set | A, B,<br>D |
| RE_TAB_F_X | 14.3.9.2 | Mean and Mean<br>Relative Change<br>from Baseline in | Safety<br>Analysis Set | A, B,<br>D |

| Rho Table Identifier <sup>a</sup> | Table No.b | Title | Population | Part |
|---|---|---|---|---|
| | | Spirometry Values<br>by Visit and Dose<br>Group | | |
| CM_TAA_F_X | 14.3.10.1 | Number and Percentage of Subjects with Concomitant Medications by Anatomic Class, Therapeutic Class, Medication Term, and Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| CM_TAB_F_X | 14.3.10.2 | Number and<br>Percentage of<br>Subjects with Prior<br>Medications by<br>Anatomic Class,<br>Therapeutic Class,<br>Medication Term<br>and Dose Group | Safety<br>Analysis Set | A, B,<br>D, O |
| QS_TAA_F_B | 14.4.1 | Mean and Mean<br>Change from<br>Baseline in CFQ-R<br>Respiratory<br>Domain Scores by<br>Visit and Dose<br>Group | Safety<br>Analysis Set | В |

<sup>&</sup>lt;sup>a</sup>The same set of tables will be produced separately for each study part, unless otherwise specified. '\_X' in each table name will reflect each study part (\_A, \_B, \_D) or overall (\_O). These tables will have the 'Dose Group' portion of the title removed.

<sup>&</sup>lt;sup>b</sup> A, B, D or O will be added to each display number.

# **15.LIST OF PLANNED FIGURES**

| Rho Figure<br>Identifier <sup>a</sup> | Figure No.b | Title | Population | Part |
|---|---|---|---|---|
| LB_FAA_F_X | 14.3.4.1.1 | C Reactive Protein (mg/L)<br>by Dose Group, Subject, and<br>Visit | Safety<br>Analysis Set | A, B, D |
| LB_FAJ_F_A | 14.3.4.1.1.1 | C Reactive Protein (mg/L)<br>by Dose Group, Subject, and<br>Visit Through Day 29 | Safety<br>Analysis Set | A |
| LB_FAJ_F_B | 14.3.4.1.1.1 | C Reactive Protein (mg/L)<br>by Dose Group, Subject, and<br>Visit Through Day 57 | Safety<br>Analysis Set | В |
| LB_FAJ_F_D | 14.3.4.1.1.1 | C Reactive Protein (mg/L)<br>by Dose Group, Subject, and<br>Visit Through Day 32 | Safety<br>Analysis Set | D |
| LB_FAB_F_X | 14.3.4.2.1 | White Blood Cells (x10^9/L) by Dose Group, Subject, and Visit | Safety<br>Analysis Set | A, B, D |
| LB_FAC_F_X | 14.3.4.3.1 | Neutrophils/Leukocytes (%) by Dose Group, Subject, and Visit | Safety<br>Analysis Set | A, B, D |
| VS_FAA_F_A | 14.3.5.1.1 | Body Temperature Values by<br>Dose Group, Subject, and<br>Visit Through Day 7 | Safety<br>Analysis Set | A |
| VS_FAA_F_B | 14.3.5.1.1 | Body Temperature Values by<br>Dose Group, Subject, and<br>Visit Through Day 36 | Safety<br>Analysis Set | В |
| VS_FAA_F_D | 14.3.5.1.1 | Body Temperature Values by<br>Dose Group, Subject, and<br>Visit Through Day 11 | Safety<br>Analysis Set | D |
| RE_FAH_F_X | 14.3.9.1.2 | Percent Predicted FEV1<br>Values by Dose Group,<br>Subject, and Visit | Safety<br>Analysis Set | A, B, D |
| RE_FAI_F_A | 14.3.9.2.2 | Percent Predicted FEV1<br>Values to Day 29 by Dose<br>Group, Subject, and Visit | Safety<br>Analysis Set | A |
| RE_FAI_F_B | 14.3.9.2.2 | Percent Predicted FEV1<br>Values to Day 57 by Dose<br>Group, Subject, and Visit | Safety<br>Analysis Set | В |

| Rho Figure<br>Identifier <sup>a</sup> | Figure No.b | Title | Population | Part |
|---|---|---|---|---|
| RE_FAI_F_D | 14.3.9.2.2 | Percent Predicted FEV1<br>Values to Day 32 by Dose<br>Group, Subject, and Visit | Safety<br>Analysis Set | D |
| RE_FAC_F_X | 14.3.9.3 | Mean and Standard Error of<br>Percent Predicted FEV1<br>Values by Dose Group and<br>Visit | Safety<br>Analysis Set | A, B, D |
| RE_FAS_F_A | 14.3.9.3.1 | Mean and Standard Error of<br>Percent Predicted FEV1<br>Values by Dose Group and<br>Visit Through Day 29 | Safety<br>Analysis Set | A |
| RE_FAS_F_B | 14.3.9.3.1 | Mean and Standard Error of<br>Percent Predicted FEV1<br>Values by Dose Group and<br>Visit Through Day 57 | Safety<br>Analysis Set | В |
| RE_FAS_F_D | 14.3.9.3.1 | Mean and Standard Error of<br>Percent Predicted FEV1<br>Values by Dose Group and<br>Visit Through Day 32 | Safety<br>Analysis Set | D |
| RE_FAL_F_X | 14.3.9.4 | Mean and Standard Error of<br>Absolute Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit | Safety<br>Analysis Set | A, B, D |
| RE_FAM_F_A | 14.3.9.4.1 | Mean and Standard Error of<br>Absolute Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 29 | Safety<br>Analysis Set | A |
| RE_FAM_F_B | 14.3.9.4.1 | Mean and Standard Error of<br>Absolute Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 57 | Safety<br>Analysis Set | В |
| RE_FAM_F_D | 14.3.9.4.1 | Mean and Standard Error of<br>Absolute Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 32 | Safety<br>Analysis Set | D |

| Rho Figure<br>Identifier <sup>a</sup> | Figure No.b | Title | Population | Part |
|---|---|---|---|---|
| RE_FAN_F_X | 14.3.9.4.2 | Mean and Standard Error of<br>Relative Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit | Safety<br>Analysis Set | A, B, D |
| RE_FAP_F_A | 14.3.9.4.3 | Mean and Standard Error of<br>Relative Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 29 | Safety<br>Analysis Set | A |
| RE_FAP_F_B | 14.3.9.4.3 | Mean and Standard Error of<br>Relative Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 57 | Safety<br>Analysis Set | В |
| RE_FAP_F_D | 14.3.9.4.3 | Mean and Standard Error of<br>Relative Change from<br>Baseline in Percent Predicted<br>FEV1 Values by Dose Group<br>and Visit to Day 32 | Safety<br>Analysis Set | D |

<sup>&</sup>lt;sup>a</sup>The same set of figures will be separately for each study part, unless otherwise specified.

<sup>&#</sup>x27;\_X' in each table name will reflect each study part (\_A, \_B, \_D).

b A, B or D will be added to each display number.

# **16.LIST OF PLANNED DATA LISTINGS**

| Rho Listing<br>Identifier <sup>a</sup> | Listing<br>No. <sup>b</sup> | Title | Population | Part |
|---|---|---|---|---|
| DS_LAA_F_X | 16.2.1.1 | Listing of Screen<br>Failures | Screened<br>Subjects | A, B, D |
| DS_LAB_F_X | 16.2.1.2 | Listing of Subject Disposition | Safety Analysis<br>Set | A, B, D |
| DS_LAC_F_X | 16.2.1.3 | Listing of Visits Not Done, Conducted as Home Health Visits, or Visits Conducted as Telephone Visits as a Replacement for a Scheduled In-Clinic Visit | Safety Analysis<br>Set | A, B, D |
| PD_LAA_F_X | 16.2.2 | Listing of Protocol Deviations | Safety Analysis<br>Set | A, B, D |
| DM_LAB_F_X | 16.2.4.1 | Listing of Demographics and Baseline Characteristics | Safety Analysis<br>Set | A, B, D |
| EX_LAB_F_B<br>EX_LAB_F_D | 16.2.5.1 | Listing of Overall Extent of Exposure | Safety Analysis<br>Set | B, D |
| EX_LAC_F_X | 16.2.5.2 | Listing of Extent of Exposure at the Visit Level | Safety Analysis<br>Set | A, B, D |
| EX_LAA_F_X | 16.2.5.3 | Listing of Investigational Product Administration | Safety Analysis<br>Set | A, B, D |
| MH_LAA_F_X | 16.2.6.1 | Listing of Medical<br>History by Subject,<br>System Organ Class, and<br>Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAA_F_X | 16.2.7.1 | Listing of Adverse<br>Events by Subject,<br>System Organ Class, and<br>Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAB_F_X | 16.2.7.2 | Listing of Adverse Events Leading to Treatment Discontinuation by Subject, System Organ | Safety Analysis<br>Set | A, B, D |

| Rho Listing<br>Identifier <sup>a</sup> | Listing<br>No.b | Title | Population | Part |
|---|---|---|---|---|
| | | Class, and Preferred<br>Term | • | |
| AE_LAD_F_X | 16.2.7.3 | Listing of Adverse<br>Events Resulting in<br>Death by Subject,<br>System Organ Class, and<br>Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAC_F_X | 16.2.7.4 | Listing of Serious<br>Adverse Events by<br>Subject, System Organ<br>Class, and Preferred<br>Term | Safety Analysis<br>Set | A, B, D |
| AE_LAL_F_X | 16.2.7.5 | Listing of Adverse<br>Events of Special Interest<br>by Subject, System<br>Organ Class, and<br>Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAF_F_X | 16.2.7.6 | Listing of Adverse Events Classified as Pulmonary Exacerbations (Investigator and Protocol-Defined) by Subject, System Organ Class, and Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAI_F_X | 16.2.7.7 | Listing of Pyrexia or<br>Elevated Body<br>Temperature Adverse<br>Events Reported During<br>and Up To 24 Hours<br>After Completion of<br>Nebulization by Subject,<br>System Organ Class, and<br>Preferred Term | Safety Analysis<br>Set | A, B, D |
| AE_LAJ_F_X | 16.2.7.8 | Listing of Adverse<br>Events Reported During<br>and Up To 24 Hours<br>After Completion of | Safety Analysis<br>Set | A, B, D |

| Rho Listing<br>Identifier <sup>a</sup> | Listing No.b | Title | Population | Part |
|---|---|---|---|---|
| | | Nebulization by Subject,<br>System Organ Class, and<br>Preferred Term | | |
| AE_LAK_F_X | 16.2.7.9 | Listing of Febrile Reactions and Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Subject and Preferred Term | Safety Analysis<br>Set | A, B, D |
| LB_LAA_F_X | 16.2.8.1 | Listing of Chemistry Values | Safety Analysis<br>Set | A, B, D |
| LB_LAB_F_X | 16.2.8.2 | Listing of Hematology<br>Values | Safety Analysis<br>Set | A, B, D |
| LB_LAC_F_X | 16.2.8.3 | Listing of Urinalysis<br>Values | Safety Analysis<br>Set | A, B, D |
| LB_LAD_F_B,<br>LB_LAD_F_D | 16.2.8.4 | Listing of Coagulation<br>Values | Safety Analysis<br>Set | B, D |
| LB_LAE_F_B<br>LB_LAE_F_D | 16.2.8.5 | Listing of Serum<br>Inflammatory Markers | Safety Analysis<br>Set | B, D |
| PG_LAA_F_X | 16.2.8.8 | Listing of Pregnancy<br>Results | Safety Analysis<br>Set | A, B, D |
| VS_LAA_F_X | 16.2.9.1 | Listing of Vital Signs | Safety Analysis<br>Set | A, B, D |
| EG_LAA_F_X | 16.2.10.1 | Listing of Overall<br>Electrocardiogram<br>Interpretation Findings | Safety Analysis<br>Set | A, B, D |
| CX_LAA_F_X | 16.2.11.1 | Listing of Chest X-Ray Findings | Safety Analysis<br>Set | A, B, D |
| PE_LAA_F_X | 16.2.12.1 | Listing of Physical Examination Results | Safety Analysis<br>Set | A, B, D |
| RE_LAA_F_X | 16.2.13.1 | Listing of Spirometry Values | Safety Analysis<br>Set | A, B, D |
| CM_LAA_F_X | 16.2.14.1 | Listing of Prior and<br>Concomitant<br>Medications | Safety Analysis<br>Set | A, B, D |

| Rho Listing<br>Identifier <sup>a</sup> | Listing<br>No. <sup>b</sup> | Title | Population | Part |
|---|---|---|---|---|
| CM_LAB_F_X | 16.2.14.2 | Listing of Concomitant<br>Surgical Procedures | Safety Analysis<br>Set | A, B, D |
| QS_LAA_F_B | 16.2.15.1 | Listing of CFQ-R<br>Respiratory Domain<br>Scores | Safety Analysis<br>Set | В |

<sup>&</sup>lt;sup>a</sup>The same set of listings will be separately for each study part, unless otherwise specified.

<sup>&#</sup>x27;\_X' in each table name will reflect each study part (\_A, \_B, \_D).

<sup>&</sup>lt;sup>b</sup>A, B or D will be added to each display number.

#### 17.APPENDICES

# 17.1 Study Flow Chart

#### Part A



## Part B



### Part D



# 17.2 Subject Enrollment and Treatment Allocation




# 17.3 Schedule of Events

The schedule of events is outlined in Table 1 through Table 9 in the protocol.

# **18.ATTACHMENTS**

- Table Display Specifications
- Listing Display Specifications
- Figure Display Specifications

# Translate Bio, Inc. PROTOCOL NUMBER MRT5005-101

A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled, Combined Single and Multiple Ascending Dose Study Evaluating the Safety, Tolerability, and Biological Activity of MRT5005 (mRNA/mr LNP) Administered by Nebulization to Adult with ic Fibrosis

# Table Specifications

VERSION DATE: 26 October 2021

SPONSOR: Translate Bio, Inc. 29 Hartwell Avenue Lexington, MA 02421 Telephone: (617) 945-7361

PREPARED BY: Rho, Inc. 2635 E NC Hwy 54 Durham, NC 27713 Telephone: (919) 408-8000 Fax: (919) 408-0999

# Table Specifications

#### Table of Contents

| Demographics |
|---|
| Table 14.1.1.1 (DM TAA F X) Summary of Demographic and Baseline Characteristics by Dose Group Population: Safety Analysis Set 6 |
| Table 14.1.1.1 (DM TAA F O) Summary of Demographic and Baseline Characteristics Population: Safety Analysis Set |
| Disposition |
| Table 14.1.3.1 (DS TAA F X) Summary of Screen Failures |
| Population: Screened Subjects |
| Table 14.1.3.2 (DS TAB F X) Summary of Subject Disposition by Dose Group Population: Safety Analysis Set |
| Treatment Compliance |
| Table 14.1.4 (EX TAA F X) Summary of Investigational Product Administration by Dose Group Population: Safety Analysis Set 12 |
| Table 14.1.4 (EX TAA F O) Summary of Investigational Product Administration Population: Safety Analysis Set |
| Medical History |
| Table 14.1.5 (MH TAA F X) Medical History by System Organ Class and Preferred Term by Dose Group Population: Safety Analysis Set 14 |
| Protocol Deviations |
| Table 14.1.6 (PD_TAA_F_X) Protocol Deviations by Type and Dose Group Population: Safety Analysis Set |
| Adverse Events |
| Table 14.3.1.1 (AE_TAA_F_X) Overall Summary of Treatment-Emergent Adverse Events by Dose Group Population: Safety Analysis Set 16 |
| Table 14.3.1.1.1 (AE_TAI_F_A) Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 29 Population: Safety |
| Analysis Set |
| Table 14.3.1.1.1 (AE_TAI_F_B) Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 57 Population: Safety |
| Analysis Set |
| Table 14.3.1.1.1 (AE_TAI_F_D) Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 32 Population: Safety |
| Analysis Set |
| Table 14.3.1.1.2 (AE_TAK_F_O) Overall Summary of Treatment-Emergent Adverse Events by Time Interval Population: Safety Analysis |
| Set |
| Table 14.3.1.2 (AE_TAB_F_X) Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Time Interval |
| and Dose Group Population: Safety Analysis Set |
| Table 14.3.2.1 (AE_TAC_F_X) Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term by Time |
| Interval and Dose Group Population: Safety Analysis Set |
| Table 14.3.2.2 (AE_TAL_F_X) Summary of Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred |
| Term by Time Interval and Dose Group Population: Safety Analysis Set |
| Table 14.3.2.3 (AE_TAE_F_X) Summary of Treatment-Emergent Adverse Events Classified as Pulmonary Exacerbations by Preferred Term by |
| Time Interval and Dose Group Population: Safety Analysis Set |
| Table 14.3.1.3 (AE_TAH_F_X) Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Population: Safety |
| Analysis Set |
| Table 14.3.1.3.1 (AE_TAJ_F_A) Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 29 |
| Population: Safety Analysis Set |
| Table 14.3.1.3.1 (AE_TAJ_F_B) Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 57 |
| Population: Safety Analysis Set |
| Table 14.3.1.3.1 (AE_TAJ_F_D) Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 32 |
| Population: Safety Analysis Set |
| Table 14.3.1.4 (AE_TAN_F_O) Number of Treatment-Emergent Adverse Events by Preferred Term and Time Interval Population: Safety |
| Analysis Set |

| Table 14.3.2.4 (AE_TAM_F_X) Summary of Treatment-Emergent Februle Reactions in First 24 Hours After Completion of Nebulization b | ıγ |
|---|---|
| Preferred Term and Dose Group Population: Safety Analysis Set | . 28 |
| Table 14.3.2.6 (AE TAP F X) Summary of Treatment-Emergent Hypersensitivity Reactions in First 24 Hours After Completion of | |
| Nebulization by Preferred Term and Dose Group Population: Safety Analysis Set | |
| Table 14.3.2.5 (AE_TAO_F_O) Summary of Treatment-Emergent Febrile Reactions in First 24 Hours After Completion of Nebulization b | у |
| Preferred Term Population: Safety Analysis Set | . 30 |
| Table 14.3.2.7 (AE_TAQ_F_0) Summary of Treatment-Emergent Hypersensitivity Reactions in First 24 Hours After Completion of | |
| Nebulization by Preferred Term Population: Safety Analysis Set | . 31 |
| Vital Signs | . 32 |
| Table 14.3.5.1 (VS_TAA_F_X) Mean and Mean Change from Baseline in Vital Signs by Visit and Dose Group Population: Safety Analy | /sis |
| Set | . 32 |
| Laboratory Values | |
| Table 14.3.4.1 (LB_TAA_F_X) Mean and Mean Change from Baseline in Chemistry Laboratory Values by Visit and Dose Group Populatio | |
| Safety Analysis Set | |
| Table 14.3.4.2 (LB_TAB_F_X) Mean and Mean Change from Baseline in Hematology Laboratory Values by Visit and Dose Group Populati | .on: |
| Safety Analysis Set | |
| Table 14.3.4.3 (LB_TAE_F_B, LB_TAE_F_D) Mean and Mean Change from Baseline in Immune Response to Serum Inflammatory Markers by | |
| Visit and Dose Group Population: Safety Analysis Set | |
| Electrocardiogram | |
| Table 14.3.6.1 (EG_TAA_F_X) Shift in Overall Electrocardiogram Interpretation Findings by Visit and Dose Group Population: Saf | |
| Analysis Set | |
| Chest X-Ray | |
| Table 14.3.7.1 (CX_TAA_F_X) Shift in Chest X-Ray by Visit and Dose Group Population: Safety Analysis Set | |
| Physical Examination | |
| Table 14.3.8.1 (PE_TAA_F_X) Summary of Physical Examination by Visit and Dose Group Population: Safety Analysis Set | |
| Spirometry | |
| Table 14.3.9.1 (RE_TAA_F_X) Mean and Mean Absolute Change from Baseline in Spirometry Values by Visit and Dose Group Population: | |
| Safety Analysis Set | |
| Table 14.3.9.2 (RE_TAB_F_X) Mean and Mean Relative Change from Baseline in Spirometry Values by Visit and Dose Group Population: | |
| Safety Analysis Set | |
| Concomitant Medications | |
| Table 14.3.10.1 (CM_TAA_F_X) Number and Percentage of Subjects with Concomitant Medications by Anatomic Class, Therapeutic Class | |
| Medication Term, and Dose Group Population: Safety Analysis Set | . 41 |
| Table 14.3.10.2 (CM_TAB_F_X) Number and Percentage of Subjects with Prior Medications by Anatomic Class, Therapeutic Class, | |
| Medication Term, and Dose Group Population: Safety Analysis Set | |
| CFQ-R | . 43 |
| Table 14.4.1 (QS_TAA_F_B) Mean and Mean Change from Baseline in CFQ-R Respiratory Domain Scores by Visit and Dose Group | |
| Population: Safety Analysis Set | . 43 |

#### General Programming Notes

The following instructions apply to all table displays.

#### DISPLAY OUTPUTS FOR EACH PART

Each table will be produced for each study part (A, B, D), unless otherwise specified. Each version of the table will include the relevant study part in the header and in the table identifier. For example, DM\_TAA\_F\_X will be identified as DM\_TAA\_F\_A for Part A and will include a header to show 'Part A'. Certain tables will also be produced for the study overall (O). For the overall tables, 'Part: All Study Parts' will print in the header and \_O will be appended to the table identifier. A, B, D or O will be added to each display number.

#### PROGRAMMER NOTES

Programmer notes appear at the bottom of each table display shell where applicable.

Dose groups for each part are as follow:

- Part A: MRT5005 8mg, MRT5005 16mg, MRT5005 20mg, MRT5005 24mg, Pooled Placebo
- Part B: MRT5005 8mg, MRT5005 12mg, MRT5005 16mg, MRT5005 20mg, Pooled Placebo
- Part D: MRT5005 4mg, Placebo

For the overall tables, the treatment groups will be Pooled MRT5005 and Pooled Placebo.

Column labels in the mock tables use MRT5005 Xmg and Pooled Placebo. For Part D tables, Placebo should be used and not Pooled Placebo.

#### PAGE FORMATTING

The specifications for the format of each page are page size=47, line size=134, font=Courier, font size=8, and margin = 1.5" top, 1" bottom, left, and right.

"Listing Source: <Listing Number>" will be printed on the right side of the footer for each table.

#### PRECISION

No preliminary rounding should be performed; rounding should only occur after analysis. To round, consider digit to right of last significant digit: if < 5 then round down, if  $\ge$  5 then round up. Means, medians, 25th percentiles, 75th percentiles, and confidence intervals will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one

Translate Bio, Inc.
Protocol No. MRT5005-101

decimal place. Minimums and maximums will be presented with the same precision as the original data, with a maximum of 4 decimal places.

## Demographics

 $\begin{tabular}{llll} Table 14.1.1.1 & (DM\_TAA\_F\_X) \\ Summary of Demographic and Baseline Characteristics by Dose Group \\ Population: Safety Analysis Set \\ \end{tabular}$ 

| Part: x | | | | |
|---|---|---|---|---|
| | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| Characteristics | N=xx | N=xx | N=xx | N=xx |
| 0.000 (0.000) | | | | |
| Sex - n (%) | , | , | , | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Age (years) [1] | | | | |
| Subject 1 | XX | XX | XX | XX |
| Subject 2 | XX | XX | XX | XX |
| Subject 3 | XX | XX | XX | XX |
| Subject 4 | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |
| Race - n (%) | | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity - n (%) | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1110011119 | AA (AA.A) | $m (M \cdot M)$ | AA (AA.A) | ΔΔ (ΔΛ•Λ) |
| Genotype - n (%) | | | | |
| Class I/Class I | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

# Translate Bio, Inc. Protocol No. MRT5005-101

| Class I/Class II | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
|---|---|---|---|---|
| Class II/Class I | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Class II/Class II | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing/xxxx | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| FTR Modulator Use at Baseline - | n (%) [2] | | | |
| Yes | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 105 | () | | | |
| No | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No ercent Predicted FEV $_1$ at Baselin | xx (xx.x) | | xx (xx.x) | |
| No ercent Predicted $FEV_1$ at Baselin 3] | xx (xx.x) ne - n (%) | xx (xx.x) | | xx (xx.x) |
| No ercent Predicted FEV $_1$ at Baselin | xx (xx.x) | | xx (xx.x)<br>xx (xx.x) | |

<sup>[1]</sup> DM F01

PC F02

Listing Source: DM LAB F X

- 1) 'Missing' row should only be included for categorical variables if there is missing data. For genotype, if only one class is missing, still display the populated mutation (i.e. Missing/Class I).
- 2) The Missing row should be included in the %s.
- 3) For Part D, replace footnote RE F01 with RE F01D.

<sup>[2]</sup> DM\_F02

<sup>[3]</sup> RE F01

AB F02

Table 14.1.1.1 (DM\_TAA\_F\_O)
Summary of Demographic and Baseline Characteristics
Population: Safety Analysis Set

| Part: All Study Parts | | |
|-------------------------------------------|----------------|----------------|
| - | Pooled MRT5005 | Pooled Placebo |
| Characteristics | N=xx | N=xx |
| | | _ |
| Sex - n (%) | | |
| Male | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) |
| Age (years) [1] | | |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Range | (xx, xx) | (xx, xx) |
| Race - n (%) | | |
| White | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) |
| Ethnicity - n (%) | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) |
| Genotype - n (%) | | |
| Class I/Class I | xx (xx.x) | xx (xx.x) |
| Class I/Class II | xx (xx.x) | xx (xx.x) |
| Class II/Class I | xx (xx.x) | xx (xx.x) |
| Class II/Class II | xx (xx.x) | xx (xx.x) |
| Missing/xxxx | xx (xx.x) | xx (xx.x) |

| Etc. | xx (xx.x) | xx (xx.x) |
|----------------------------------------------------|-----------|-----------|
| CFTR Modulator Use at Baseline - n (%) [2] | | |
| Yes | xx (xx.x) | xx (xx.x) |
| No | xx (xx.x) | xx (xx.x) |
| Percent Predicted $FEV_1$ at Baseline - n (%) [3] | | |
| < 70 | xx (xx.x) | xx (xx.x) |
| ≥ 70 | xx (xx.x) | xx (xx.x) |
| Percent Predicted FEV <sub>1</sub> at Baseline [3] | | |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Range | (xx, xx) | (xx, xx) |

PC F02

Listing Source: DM\_LAB\_F\_X

- 1) 'Missing' row should only be included for categorical variables if there is missing data. For genotype, if only one class is missing, still display the populated mutation (i.e. Missing/Class I).
- 2) The Missing row should be included in the %s.

<sup>[1]</sup> DM F01

<sup>[2]</sup> DM F02

<sup>[3]</sup> RE F010

AB F02

## Disposition

Table 14.1.3.1 (DS\_TAA\_F\_X) Summary of Screen Failures Population: Screened Subjects

| | Total |
|---------------------------|-----------|
| | N=xx |
| | n (%) |
| Screened | xx |
| Screen failure | xx (xx.x) |
| Randomized | xx (xx.x) |
| Reason for screen failure | |
| Adverse Event | |
| Inclusion/exclusion | xx (xx.x) |
| Lost to follow-up | xx (xx.x) |
| Withdrew consent | xx (xx.x) |
| Other | xx (xx.x) |

Note: PC F02

Listing Source: DS\_LAA\_F\_X

- 1) Please check footnotes for denominators.
- 2) DS\_TAA\_F\_X will be produced for each study part and for the study overall.

Table 14.1.3.2 (DS\_TAB\_F\_X)
Summary of Subject Disposition by Dose Group
Population: Safety Analysis Set

| Part: x | | | | |
|---|---|---|---|---|
| | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| | N=xx | N=xx | N=xx | N=xx |
| | n (%) | n (%) | n (%) | n (%) |
| Study completion status [1] | | | | |
| Completed | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for premature study | | | | |
| discontinuation [2] | | | | |
| Adverse event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Study terminated by sponsor | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> PC\_F02

Listing Source: DS LAB F X

- 1) Please check footnotes for denominators.
- 2) DS\_TAB\_F\_X will be produced for each study part and for the study overall.

<sup>[2]</sup> DS\_F03

#### Treatment Compliance

Table 14.1.4 (EX\_TAA\_F\_X)

Summary of Investigational Product Administration by Dose Group
Population: Safety Analysis Set

| Part: x | | | | |
|---|---|---|---|---|
| | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| | N=xx | N=xx | N=XX | N=xx |
| Number of Total Doses Administered | 1 - n | | | |
| (%) | , | , | | |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Full Doses Administered | | | | |
| Subject 1 | XX | xx | xx | XX |
| Subject 2 | XX | xx | xx | XX |
| Subject 3 | XX | xx | xx | xx |
| Subject 4 | XX | xx | xx | xx |
| Mean | XX.X | xx.x | xx.x | xx.x |
| SD | xx.xx | XX.XX | XX.XX | XX.XX |
| Number of Partial Doses Administer | red | | | |
| Subject 1 | XX | XX | XX | XX |
| Subject 2 | XX | xx | XX | XX |
| Subject 3 | XX | XX | XX | xx |
| Subject 4 | XX | XX | XX | xx |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD | XX.XX | XX.XX | XX.XX | XX.XX |

AB\_F01a PC\_F02 EX F01

Listing Source: EX\_LAB\_F\_X, EX\_LAC\_F\_X

#### Notes:

1) For Part A, only display the category for 1 Total Dose Administered, and do not present the summary statistics. For Parts B and D, please display all categories for number of doses administered (1-5) and summary statistics. The number of doses section is the sum of full and partial doses.

Table 14.1.4 (EX\_TAA\_F\_O)
Summary of Investigational Product Administration
Population: Safety Analysis Set

| Part: All Study Parts | Pooled MRT5005<br>N=xx | Pooled Placebo<br>N=xx |
|---|---|---|
| Number of Total Doses Administered - n (%) | | |
| 1 | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) |
| Number of Full Doses Administered | | |
| Mean | XX.X | XX.X |
| SD | XX.XX | XX.XX |
| Range | (xx, xx) | (xx, xx) |
| Number of Partial Doses Administered | | |
| Mean | XX.X | xx.x |
| SD | xx.xx | xx.xx |
| Range | (xx, xx) | (xx, xx) |

AB\_F01 PC\_F02 EX\_F01

Listing Source: EX\_LAB\_F\_X, EX\_LAC\_F\_X

#### Medical History

Table 14.1.5 (MH\_TAA\_F\_X)

Medical History by System Organ Class and Preferred Term by Dose Group
Population: Safety Analysis Set

| Part: x | | | | |
|---|---|---|---|---|
| | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| System Organ Class | N=xx | N=xx | N=XX | N=xx |
| Preferred Term | n (%) | n (%) | n (%) | n (%) |
| Any Medical History | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

PC\_F02 MH F01

Listing Source: MH LAA F X

- 1) MH\_TAA\_F\_X will be produced for each study part and for the study overall.
- 2) Sort System Organ Class and Preferred Term within System Organ Class by descending order of overall (MRT5005 + Placebo) frequency.

#### Protocol Deviations

# Table 14.1.6 (PD\_TAA\_F\_X) Protocol Deviations by Type and Dose Group Population: Safety Analysis Set

| Part: x | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
|---|---|---|---|---|
| Type | N=xx<br>n (%) | N=xx<br>n (%) | N=xx<br>n (%) | N=xx<br>n (%) |
| 1750 | 11 (0) | 11 (0) | 11 (0) | 11 (0) |
| Any Protocol Deviation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Type 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

PC F02

Listing Source: PD LAA F X

- 1) PD TAA F X will be produced for each study part.
- 2) Sort Type by descending order of overall (MRT5005 + Placebo) frequency.

#### Adverse Events

Table 14.3.1.1 (AE\_TAA\_F\_X)

Overall Summary of Treatment-Emergent Adverse Events by Dose Group

Population: Safety Analysis Set

| Part: x | MRT5005 Xr<br>N=xx | 3 | 5005 Xmg<br>N=xx | | 5005 Xmg<br>N=xx | | d Placebo<br>N=xx |
|---|---|---|---|---|---|---|---|
| | n (%) | | n (%) | 1 | ૧ (%) | ľ | n (%) |
| Number of TEAEs Reported | xx | | xx | | XX | | XX |
| Number of Subjects with Any TEAE Reported [1] | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Number of Serious TEAEs Reported | xx | | XX | | XX | | xx |
| Number of Subjects with Any Serious TEAE Reported [1] | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Number of TEAEs by Relationship to IP | | | | | | | |
| Not Related | XX | | XX | | XX | | XX |
| Related | XX | | XX | | XX | | XX |
| Number of Subjects with TEAEs by Relationship to IP [2] | | | | | | | |
| Not Related | xx (xx.x) | | (xx.x) | | (xx.x) | XX | (xx.x) |
| Related | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs by Relationship to Nebulization/Treatment Administration [3] | | | | | | | |
| Not Related | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Related | xx (xx.x) | xx | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Number of TEAEs by Severity | | | | | | | |
| Mild | XX | | XX | | XX | | XX |
| Moderate | XX | | XX | | XX | | XX |
| Severe | XX | | XX | | XX | | XX |
| Number of Subjects with TEAEs by Severity [4] | | | | | | | |
| Mild | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Moderate | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Severe | xx (xx.x) | XX | (xx.x) | XX | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs Leading to Treatment Discontinuation [1] | xx (xx.x) | xx | (xx.x) | xx | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs Resulting in Death [1] | xx (xx.x) | xx | (xx.x) | XX | (xx.x) | xx | (xx.x) |
| Number of TEAEs Classified as a Pulmonary Exacerbation by Type | | | | | | | |
| All | xx | | xx | | xx | | xx |

| Investigator-Defined | XX | xx | XX | XX |
|---|---|---|---|---|
| Protocol-Defined | XX | XX | XX | XX |
| Number of Subjects with TEAEs Classified as a Pulmonary | | | | |
| Exacerbation by Type [1] | | | | |
| All [5] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator-Defined | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Protocol-Defined | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

AB F03

- [1] AE F05
- [2] AE F06a
- [3] AE F06b
- [4] AE F07
- [5] AE F06d
- PC F02

Listing Source: AE LAA F X

- 1) The rows 'Number of TEAEs Reported' and 'Number of Serious TEAEs Reported' display the total number of TEAE counts.
- 2) If a subject experiences multiple adverse events, then take the closest relationship to study drug for the row 'Number of Subjects with TEAEs by Relationship' for each relationship to IP and relationship to nebulization
- 3) If a subject experiences multiple adverse events, then take the worst case severity for the row 'Number of Subjects with TEAES by Severity'.
- 4) In the by type summary of subjects with TEAEs classified as pulmonary exacerbations, any subject with either investigator-defined or protocol-defined will be counted once in the All row. Subjects with both an investigator-defined and a protocol-defined TEAE classified as a pulmonary exacerbation will be recorded once in each row, investigator-defined and protocol-defined.

```
Non-unique tables for AE_TAA_F_X:
                                                     Table 14.3.1.1.1 (AE TAI F A)
                           Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 29
                                                   Population: Safety Analysis Set
AB F03
[1] AE F05
[2] AE F06a
[3] AE F06b
[4] AE F07
[5] AE F06d
PC F02
Listing Source: AE LAA F A
                                                     Table 14.3.1.1.1 (AE TAI F B)
                           Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 57
                                                   Population: Safety Analysis Set
AB F03
[1] AE F05
[2] AE F06a
[3] AE F06b
[4] AE F07
[5] AE F06d
PC F02
Listing Source: AE LAA F B
                                                     Table 14.3.1.1.1 (AE TAI F D)
                           Overall Summary of Treatment-Emergent Adverse Events by Dose Group Through Day 32
                                                   Population: Safety Analysis Set
AB F03
[1] AE F05
[2] AE F06a
[3] AE F06b
[4] AE F07
[5] AE F06d
PC F02
```

Listing Source: AE LAA F D

Table 14.3.1.1.2 (AE\_TAK\_F\_O)

Overall Summary of Treatment-Emergent Adverse Events by Time Interval Population: Safety Analysis Set

| | Pooled MRT5005<br>N=xx | | Pooled Placebo<br>N=xx | |
|---|---|---|---|---|
| | r | 1 (%) | r | n (%) |
| Viniban of BENES Demonted | | | | |
| Number of TEAEs Reported | | XX | | XX |
| Number of Subjects with Any TEAE Reported [1] | XX | (xx.x) | XX | (xx.x) |
| Number of Serious TEAEs Reported | | XX | | XX |
| Number of Subjects with Any Serious TEAE Reported [1] | XX | (xx.x) | XX | (xx.x) |
| Number of TEAEs by Relationship to IP | | | | |
| Not Related | | XX | | XX |
| Related | | XX | | XX |
| Number of Subjects with TEAEs by Relationship to IP [2] | | | | |
| Not Related | XX | (xx.x) | XX | (xx.x) |
| Related | XX | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs by Relationship to<br>Nebulization/Treatment Administration [3] | | | | |
| Not Related | ×× | (xx.x) | vv | (xx.x) |
| Related | | (xx.x) | | (xx.x) |
| Number of TEAEs by Severity | | | | |
| Mild | | XX | | XX |
| Moderate | | XX | | XX |
| Severe | | XX | | XX |
| Number of Subjects with TEAEs by Severity [4] | | | | |
| Mild | XX | (xx.x) | XX | (xx.x) |
| Moderate | XX | (xx.x) | XX | (xx.x) |
| Severe | XX | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs Leading to Treatment<br>Discontinuation [1] | XX | (xx.x) | XX | (xx.x) |
| Number of Subjects with TEAEs Resulting in Death [1] | XX | (xx.x) | XX | (xx.x) |
| Number of TEAEs Classified as a Pulmonary Exacerbation | | | | |
| by Type All | | xx | | XX |
| Investigator-Defined | | XX | | XX |

| Protocol-Defined | XX | xx |
|---|---|---|
| Number of Subjects with TEAEs Classified as a Pulmonary | | |
| Exacerbation by Type [1] | | |
| All [5] | xx (xx.x) | xx (xx.x) |
| Investigator-Defined | xx (xx.x) | xx (xx.x) |
| Protocol-Defined | xx (xx.x) | xx (xx.x) |

AB F03 [1] AE F05

[2] AE F06a

[3] AE F06b

[4] AE F07

[5] AE F06d PC F02

AE F18

Listing Source: AE LAA F X

- 1) The first page will be "Part: All Study Parts" with "Time Interval: Overall" and will include all AEs across all study parts. The subsequent page will be: "Part: All Study Parts" with "Time Interval: 1 month post-dose". The last page will be: "Part: All Study Parts" with "Time Interval: > 1 month post-dose".
- 2) In the column headers, report the number of subjects who were at risk for an AE at the start of the interval.
- 3) The rows 'Number of TEAEs Reported' and 'Number of Serious TEAEs Reported' display the total number of TEAE counts.
- 4) If a subject experiences multiple adverse events, then take the closest relationship to study drug for the row 'Number of Subjects with TEAEs by Relationship' for each relationship to IP and relationship to nebulization
- 5) If a subject experiences multiple adverse events, then take the worst case severity for the row 'Number of Subjects with TEAEs
- 6) In the by type summary of subjects with TEAEs classified as pulmonary exacerbations, any subject with either investigatordefined or protocol-defined will be counted once in the All row. Subjects with both an investigator-defined and a protocoldefined TEAE classified as a pulmonary exacerbation will be recorded once in each row, investigator-defined and protocoldefined.

Table 14.3.1.2 (AE\_TAB\_F\_X)

Summary of Treatment-Emergent Adverse Events by System Organ Class and Preferred Term by Time Interval and Dose Group Population: Safety Analysis Set

| Part: x | | | | |
|---|---|---|---|---|
| Time Interval: xx to xx | | | | |
| | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| System Organ Class | N=xx | N=xx | N=xx N=xx | |
| Preferred Term | n (%) m | n (%) m | n (%) m | n (%) m |
| System Organ Class 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

AB\_F04 AE\_F08 AE\_F14

AE\_F14 AE F15

AE F16

Listing Source: AE LAA F X

- 1) Repeat for each time interval. Time intervals for Part A are Overall, Study Day 1, 1 < Study Day  $\leq$  7, 1  $\leq$  Study Day  $\leq$  29, Study Day > 29. Time intervals for Part B are Overall, Study Day 1, 1 < Study Day  $\leq$  7, 1  $\leq$  Study Day  $\leq$  36, 1  $\leq$  Study Day  $\leq$  57, and Study Day > 57. Time intervals for Part D are Overall, Study Day 1, 1 < Study Day  $\leq$  5, 1  $\leq$  Study Day  $\leq$  11, 1  $\leq$  Study Day  $\leq$  32, and Study Day > 32.
- 2) In the column headers, report the number of subjects who were at risk for an AE at the start of the interval.
- 3) Sort System Organ Class and Preferred Term within System Organ Class by descending order of overall (MRT5005 + Placebo) frequency in subject counts.
- 4) The number of events will be summarized such that subjects with multiple TEAEs in system organ class in a time interval are counted more than once. Subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

Translate Bio, Inc.
Protocol No. MRT5005-101

#### Non-unique tables for AE\_TAB\_F\_X:

Table 14.3.2.1 (AE TAC F X)

Summary of Treatment-Emergent Serious Adverse Events by System Organ Class and Preferred Term by Time Interval and Dose Group
Population: Safety Analysis Set

AB\_F04 AE\_F08 AE\_F14 AE\_F15 AE\_F16

Listing Source: AE LAC F X

#### Notes:

- 1) AE\_TAC\_F\_X will be provided for each study part.
- 2) Repeat AE\_TAB\_F\_X for Serious Adverse Events.

Table 14.3.2.2 (AE TAL F X)

Summary of Treatment-Emergent Adverse Events of Special Interest by System Organ Class and Preferred Term by Time Interval and Dose Group

Population: Safety Analysis Set

AB\_F04 AE\_F08 AE\_F14 AE\_F15 AE\_F16

Listing Source: AE LAL F X

- 1) AE TAL F X will be provided for each study part.
- 2) Repeat AE TAB F X for AESIs.
Table 14.3.2.3 (AE TAE F X)

Summary of Treatment-Emergent Adverse Events Classified as Pulmonary Exacerbations by Preferred Term by Time Interval and Dose Group

Population: Safety Analysis Set

| Part: x<br>Time Interval: xx to xx | | | | |
|---|---|---|---|---|
| Preferred Term | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| Type | N=xx | N=xx | N=xx | N=xx |
| | n (%) m | n (%) m | n (%) m | n (%) m |
| Preferred Term 1 | | | | |
| All | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Investigator-Defined | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Protocol-Defined | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | | | | |
| All | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Investigator-Defined | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Protocol-Defined | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |

AB\_F04

AE F09

AE F14a

AE F15

AE F16

Listing Source: AE LAF F X

- 1) Repeat for each time interval. Time intervals for Part A are Overall, Study Day 1, 1 < Study Day ≤ 7, 1 ≤ Study Day ≤ 29, Study Day > 29. Time intervals for Part B are Overall, Study Day 1, 1 < Study Day ≤ 7, 1 ≤ Study Day ≤ 36, 1 ≤ Study Day ≤ 57, and Study Day > 57. Time intervals for Part D are Overall, Study Day 1, 1 < Study Day ≤ 5, 1 ≤ Study Day ≤ 11, 1 ≤ Study Day ≤ 32, and Study Day > 32.
- 2) In the column headers, report the number of subjects who were at risk for an AE at the start of the interval.
- 3) Report pulmonary exacerbations by type (all, investigator-defined and protocol-defined).
- 4) Sort Preferred Term by descending order of overall (MRT5005 + Placebo) frequency in subject counts.
- 5) The number of events will be summarized such that subjects with multiple TEAEs in a preferred term in a time interval in a type are counted more than once.

| Part: x | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
|------------------|-------------|-------------|-------------|----------------|
| | N=xx | N=xx | N=xx | N=xx |
| Preferred Term | Events | Events | Events | Events |
| | 200000 | 2.00.00 | 2.0 | 2101100 |
| Preferred Term 1 | XX | XX | XX | XX |
| Preferred Term 2 | XX | XX | XX | XX |
| Preferred Term 3 | XX | XX | XX | XX |
| Etc. | | | | |

AB\_F04 AE\_F09 AE\_F14a

AE F19

Listing Source: AE LAA F X

#### Notes:

- 1) Sort by descending order of overall (MRT5005 + Placebo) frequency.
- 2) Summarize number of events, so subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

Table 14.3.1.3.1 (AE\_TAJ\_F\_A)

Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 29

Population: Safety Analysis Set

| Part: x | | | | | |
|---|---|---|---|---|---|
| | MRT5005 8mg | MRT5005 16mg | MRT5005 20mg | MRT5005 24mg | Pooled Placebo |
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| Preferred Term | Events | Events | Events | Events | Events |
| Preferred Term 1 | XX | XX | XX | XX | XX |
| Preferred Term 2 | XX | XX | XX | XX | xx |
| Preferred Term 3 | XX | xx | XX | XX | XX |
| Etc. | | | | | |

AB\_F04 AE F09

AE\_F14a

AE F19

Listing Source: AE LAA F A

#### Notes:

- 1) Sort by descending order of overall (MRT5005 + Placebo) frequency.
- 2) Summarize number of events, so subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

#### Table 14.3.1.3.1 (AE TAJ F B)

Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 57
Population: Safety Analysis Set

| Part: x | | | | | |
|---|---|---|---|---|---|
| | MRT5005 8mg | MRT5005 12mg | MRT5005 16mg | MRT5005 20mg | Pooled Placebo |
| | N=xx | N=xx | N=xx | N=xx | N=xx |
| Preferred Term | Events | Events | Events | Events | Events |
| Preferred Term 1 | XX | XX | XX | XX | XX |
| Preferred Term 2 | xx | xx | xx | xx | xx |
| Preferred Term 3 | xx | XX | xx | xx | XX |
| Etc. | | | | | |

AB\_F04 AE F09

AE F14a

AE F19

Listing Source: AE LAA F B

#### Notes:

- 1) Sort by descending order of overall (MRT5005 + Placebo) frequency.
- 2) Summarize number of events, so subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

Table 14.3.1.3.1 (AE TAJ F D)

Number of Treatment-Emergent Adverse Events by Preferred Term by Dose Group Through Day 32 Population: Safety Analysis Set

| Part: x | | |
|------------------|-------------|---------|
| | MRT5005 4mg | Placebo |
| | N=xx | N=xx |
| Preferred Term | Events | Events |
| Preferred Term 1 | XX | XX |
| Preferred Term 2 | xx | XX |
| Preferred Term 3 | xx | XX |
| Etc. | | |

AB F04

AE\_F09 AE\_F14a AE\_F19

Listing Source: AE\_LAA\_F\_D

- 1) Sort by descending order of overall (MRT5005 + Placebo) frequency.
- 2) Summarize number of events, so subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

| Part: x Time Interval: x | | |
|--------------------------|----------------|----------------|
| | Pooled MRT5005 | Pooled Placebo |
| | N=xx | N=xx |
| Preferred Term | Events | Events |
| Preferred Term 1 | XX | xx |
| Preferred Term 2 | XX | xx |
| Preferred Term 3 | XX | xx |
| Etc. | | |

AB\_F04 AE\_F09 AE\_F14a AE\_F19 AE\_F18

- 1) The first page will be "Part: All Study Parts" with "Time Interval: Overall" and will include all AEs across all study parts. The subsequent page will be: "Part: All Study Parts" with "Time Interval: 1 month post-dose"
- 2) In the column headers, report the number of subjects who were at risk for an AE at the start of the interval.
- 3) Sort by descending order of overall (Pooled MRT5005 + Pooled Placebo) frequency.
- 4) Summarize number of events, so subjects with multiple TEAEs in preferred term in a time interval are counted more than once.

Table 14.3.2.4 (AE\_TAM\_F\_X)

Summary of Treatment-Emergent Febrile Reactions in First 24 Hours After Completion of Nebulization by Preferred Term and Dose Group Population: Safety Analysis Set

| | MRT5005 Xmg<br>N=xx<br>n (%) | MRT5005 Xmg<br>N=xx<br>n (%) | MRT5005 Xmg<br>N=xx<br>n (%) | Pooled Placebo<br>N=xx<br>n (%) |
|---|---|---|---|---|
| Number of Febrile Reactions Reported | XX | XX | XX | XX |
| Number of Subjects with Any Febrile Reactions Reported [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Febrile Reactions by Severity [2] | | | | |
| Mild | XX | XX | XX | XX |
| Moderate | xx | XX | XX | XX |
| Severe | XX | XX | XX | xx |
| Number of Subjects with Febrile Reactions by Maximum Severity [3] | | | | |
| Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

<sup>[1]</sup> AE F05

Note: AE F17a

Listing Source: AE LAK F X

#### Notes:

1) AE\_TAM\_F\_X will be produced for each study part.

<sup>[2]</sup> AE F17c

<sup>[3]</sup> AE\_F07a

Table 14.3.2.6 (AE\_TAP\_F\_X)

Summary of Treatment-Emergent Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Preferred Term and Dose Group

Population: Safety Analysis Set

| | MRT5005 Xmg<br>N=xx | MRT5005 Xmg<br>N=xx | MRT5005 Xmg<br>N=xx | Pooled Placebo<br>N=xx |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| Number of Hypersensitivity Reactions Reported | XX | XX | XX | XX |
| Number of Subjects with Any Hypersensitivity Reactions Reported [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Hypersensitivity Reactions by Severity | | | | |
| Mild | XX | XX | XX | xx |
| Moderate | XX | XX | XX | XX |
| Severe | XX | XX | XX | XX |
| Number of Subjects with Hypersensitivity Reactions by Maximum Severity | | | | |
| [2] | | | | |
| Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

[1] AE F05

[2] AE\_F07b

Note: AE F17b

Listing Source: AE LAK F X

#### Notes:

1) AE\_TAM\_F\_X will be produced for each study part.

Table 14.3.2.5 (AE\_TAO\_F\_O)

Summary of Treatment-Emergent Febrile Reactions in First 24 Hours After Completion of Nebulization by Preferred Term Population: Safety Analysis Set

| | Pooled MRT5005<br>N=xx<br>n (%) | | Pooled Place<br>N=xx<br>n (%) | |
|---|---|---|---|---|
| Number of Febrile Reactions Reported | | XX | | xx |
| Number of Subjects with Any Febrile Reactions Reported [1] | XX | (xx.x) | XX | (xx.x) |
| Number of Febrile Reactions by Severity [2] | | | | |
| Mild | | XX | | XX |
| Moderate | | XX | | XX |
| Severe | | XX | | XX |
| Number of Subjects with Febrile Reactions by Maximum Severity [3] | | | | |
| Mild | XX | (xx.x) | XX | (xx.x) |
| Moderate | XX | (xx.x) | XX | (xx.x) |
| Severe | XX | (xx.x) | XX | (xx.x) |

<sup>[1]</sup> AE F05

Note: AE F17a

Listing Source: AE\_LAK\_F\_X

<sup>[2]</sup> AE F17c

<sup>[3]</sup> AE F07a

Table 14.3.2.7 (AE\_TAQ\_F\_O)

Summary of Treatment-Emergent Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Preferred Term Population: Safety Analysis Set

| | Pooled MRT5005<br>N=xx<br>n (%) | Pooled Placebo<br>N=xx<br>n (%) |
|---|---|---|
| Number of Hypersensitivity Reactions Reported | XX | xx |
| Number of Subjects with Any Hypersensitivity Reactions Reported [1] | xx (xx.x) | xx (xx.x) |
| Number of Hypersensitivity Reactions by Severity | | |
| Mild | xx | XX |
| Moderate | XX | XX |
| Severe | XX | xx |
| Number of Subjects with Hypersensitivity Reactions by Maximum Severity [2] | | |
| Mild | xx (xx.x) | xx (xx.x) |
| Moderate | xx (xx.x) | xx (xx.x) |
| Severe | xx (xx.x) | xx (xx.x) |

[1] AE\_F05 [2] AE F07b

Note: AE\_F17b

Listing Source: AE\_LAK\_F\_X

#### Vital Signs

Table 14.3.5.1 (VS\_TAA\_F\_X)

Mean and Mean Change from Baseline in Vital Signs by Visit and Dose Group
Population: Safety Analysis Set

| Part: x | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | MRT5005 Xmg | | MRT50 | 005 Xmg | MRT5 | 005 Xmg | Poole | d Placebo |
| Parameter (unit) | 1 | N=xx | N | =xx | 1 | I=xx | | N=xx |
| Visit<br>Statistic | Actual | Absolute<br>Change from<br>Baseline | Actual | Absolute<br>Change<br>from<br>Baseline | Actual | Absolute<br>Change from<br>Baseline | Actual | Absolute<br>Change from<br>Baseline |
| Parameter 1 (unit)<br>Baseline | | | | | | | | |
| Subject 1 | XX | | XX | | xx | | XX | |
| Subject 2 | XX | | XX | | XX | | XX | |
| Subject 3 | XX | | XX | | XX | | XX | |
| Subject 4 | XX | | XX | | XX | | XX | |
| Mean | XX.X | | XX.X | | XX.X | | xx.x | |
| SD | xx.xx | | XX.XX | | XX.XX | | XX.XX | |
| DAY 1 (0HRPOST-DOSE) | | | | | | | | |
| Subject 1 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 2 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 3 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Etc. | | | | | | | | |

AB\_F01a

BL F01

CH F01

VS F01 (for Parts A and B)

Listing Source: VS LAA F X

- 1) Parameters include: Systolic Blood Pressure, Diastolic Blood Pressure, Pulse Rate, Respiratory Rate, Temperature, Height, Weight, BMI, Pulse Oximetry.
- 2) Include all post-baseline visits/timepoints where vital signs are collected for Systolic Blood Pressure, Diastolic Blood Pressure, Pulse Rate, Respiratory Rate, Temperature, Weight, Pulse Oximetry.
- 3) For any parameter collected multiple times during the nebulization period, select the latest 'DOSING' record for that dosing day.
- 4) Include baseline only for Height and BMI.
- 5) Exclude Part A Day 1 (Dosing) records.

```
Translate Bio, Inc.
Protocol No. MRT5005-101
```

#### Laboratory Values

Non-unique tables for VS\_TAA\_F\_X:

Table 14.3.4.1 (LB TAA F X)

Mean and Mean Change from Baseline in Chemistry Laboratory Values by Visit and Dose Group

Population: Safety Analysis Set

AB\_F01a BL\_F01 CH F01

Listing Source: LB LAA F X

#### Notes:

- 1) Parameters include: all chemistry laboratory test names, excluding beta-human chorionic gonadotropin
- 2) Include all visits where chemistry laboratory tests are collected.

Table 14.3.4.2 (LB TAB F X)

Mean and Mean Change from Baseline in Hematology Laboratory Values by Visit and Dose Group
Population: Safety Analysis Set

AB\_F01a BL\_F01 CH\_F01

Listing Source: LB LAB F X

#### Notes:

- 1) Parameters include: all hematology laboratory test names, excluding mean corpuscular hemoglobin and mean platelet volume.
- 2) Include all visits where hematology laboratory tests are collected.

Table 14.3.4.3 (LB\_TAE\_F\_B, LB\_TAE\_F\_D)

Mean and Mean Change from Baseline in Immune Response to Serum Inflammatory Markers by Visit and Dose Group Population: Safety Analysis Set

AB\_F01a BL\_F01 CH F01

Listing Source: LB LAG F B, LB LAG F D

- 1) Parameters include: all inflammatory marker
- 2) Include all visits where inflammatory markers are collected.

#### Electrocardiogram

Table 14.3.6.1 (EG\_TAA\_F\_X)

Shift in Overall Electrocardiogram Interpretation Findings by Visit and Dose Group
Population: Safety Analysis Set

| Part x | | | | | | Base | eline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | MRT5005 Xmg<br>N=xx | | | MRT5005 Xm | g | | MRT5005 Xm | g | Pooled Placebo<br>N=xx | | |
| | Normal | Abnormal,<br>NCS | Abnormal,<br>CS | Normal | Abnormal,<br>NCS | Abnormal,<br>CS | Normal | Abnormal,<br>NCS | Abnormal,<br>CS | Normal | Abnormal,<br>NCS | Abnormal,<br>CS |
| Visit<br>Result | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) | nn<br>n (%) |
| DAY 1<br>(Pre-dose)<br>Normal | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) |
| Abnormal,<br>NCS | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx<br>(xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal,<br>CS | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| DAY 1 (8<br>HOURS<br>POSTDOSE)<br>Normal | nn<br>xx(xx.x) | nn<br>xx (xx.x) | nn<br>xx (xx.x) | nn<br>xx(xx.x) | nn<br>xx (xx.x) | nn<br>xx (xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) | nn<br>xx<br>(xx.x) | nn<br>xx(xx.x) | nn<br>xx(xx.x) |
| Abnormal, | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx (xx.x) | xx (xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Abnormal,<br>CS | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) | xx(xx.x) |
| Etc. | | | | | | | | | | | | |

AB\_F05 VIS\_F01

EG\_F02 (for Parts A and B) or EG\_F01D for Part D EG\_F01 Listing Source: EG LAA F  $\rm X$ 

- 1) Include all visits where ECGs were scheduled per the protocol.
- 2) Only subjects with non-missing values at baseline and the post-baseline visit are included in the denominators for the percentages.

#### Chest X-Ray

Non-unique tables for  $EG\_TAA\_F\_X$ :

Table 14.3.7.1 (CX\_TAA\_F\_X)

Shift in Chest X-Ray by Visit and Dose Group
Population: Safety Analysis Set

AB\_F05 VIS\_F01 BL\_F01 XR\_F01

Listing Source:  $CX_LAA_F_X$ 

- 1) Include all visits where chest x-ray was scheduled per the protocol.
- 2) Only subjects with non-missing values at baseline and the post-baseline visit are included in the denominators for the percentages.

#### Physical Examination

### Table 14.3.8.1 (PE\_TAA\_F\_X) Summary of Physical Examination by Visit and Dose Group Population: Safety Analysis Set

| Part: x | | | | |
|---|---|---|---|---|
| Parameter | MRT5005 Xmg | MRT5005 Xmg | MRT5005 Xmg | Pooled Placebo |
| Visit | N=xx | N=xx | N=xx | N=xx |
| Result | n/nn (%) | n/nn (%) | n/nn (%) | n/nn (%) |
| General Appearance | | | | |
| Baseline | | | | |
| Normal | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx ( $xx.x$ ) | xx/xx (xx.x) |
| Abnormal, Not Clinically Significant | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) |
| Abnormal, Clinically Significant | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) |
| DAY 1 | | | | |
| Normal | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx ( $xx.x$ ) |
| Abnormal, Not Clinically Significant | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) |
| Abnormal, Clinically Significant | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) | xx/xx (xx.x) |

BL\_F01S  $\overline{\mbox{(for Parts A and B); BL_F01P}}$  (for Part D) VIS\_F01a

Listing Source: PE LAA F X

- 1) Include all visits where physical examination was done.
- 2) Include all physical examination parameters
- 3) Only subject with non-missing values at each visit are included in the denominators for the percentages.
- 4) For Part D, label Screening as Baseline

#### Spirometry

| Part: x | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | MRT5 | 005 Xmg | MRT5 | 005 Xmg | MRT5 | 005 Xmg | Poole | d Placebo |
| Parameter (unit) | I | N=xx | N=xx | | N=xx | | N=xx | |
| Visit<br>Statistic | Actual | Absolute<br>Change from<br>Baseline | Actual | Absolute<br>Change from<br>Baseline | Actual | Absolute<br>Change from<br>Baseline | Actual | Absolute<br>Change from<br>Baseline |
| Parameter 1 (unit) | | | | | | | | |
| Baseline [1] | | | | | | | | |
| Subject 1 | XX | | XX | | XX | | XX.X | |
| Subject 2 | XX | | XX | | XX | | XX.XX | |
| Subject 3 | XX | | XX | | XX | | XX | |
| Subject 4 | XX | | XX | | XX | | XX | |
| Mean | XX.X | | XX.X | | xx.x | | XX | |
| SD | xx.xx | | XX.XX | | xx.xx | | XX | |
| SE | XX.XX | | XX.XX | | XX.XX | | XX | |
| Day 1 (8 HOURS<br>POSTDOSE) | | | | | | | | |
| Subject 1 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 2 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 3 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | xx.x | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| SE | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX | XX.XX |
| Etc. | | | | | | | | |

AB F01

[1] RE\_F01 (Parts A and B) and RE\_F01D (Part D)

CH F01

Listing Source: RE\_LAA\_F\_X

#### Notes:

- 1) Parameters include: FEV1, Percent Predicted FEV1, FVC, Percent Predicted FVC, FEV1/FVC, FEF25-75%, PEF
- 2) Include all planned (per the protocol) post-baseline visits/timepoints where spirometry is performed and collected.

Non-unique tables for RE\_TAA\_F\_X:

Table 14.3.9.2 (RE TAB F X)

Mean and Mean Relative Change from Baseline in Spirometry Values by Visit and Dose Group
Population: Safety Analysis Set

AB F01

[1] RE\_F01 (Parts A and B) and RE\_F01D (Part D)

Listing Source: RE LAA F X

- 1) Repeat table RE TAA F X and summarize relative change from baseline rather than absolute change from baseline.
- 2) Replace "Absolute" in column headers with "Relative".

#### Concomitant Medications

Table 14.3.10.1 (CM TAA F X)

Number and Percentage of Subjects with Concomitant Medications by Anatomic Class, Therapeutic Class, Medication Term, and Dose Group Population: Safety Analysis Set

| Part: x Anatomic Class Therapeutic Class Medication Term | MRT5005 Xmg<br>N=xx<br>n (%) | MRT5005 Xmg<br>N=xx<br>n (%) | MRT5005 Xmg<br>N=xx<br>n (%) | Total<br>N=xx<br>n (%) |
|---|---|---|---|---|
| redicación feim | 11 (0) | 11 (0) | 11 (0) | 11 (0) |
| Any Concomitant Medication | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anatomic Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Anatomic Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Therapeutic Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Etc.

CM F01 CM F02

CM F03

CM F04

CM F05

CM F06 CM F08

Listing Source: CM\_LAA\_F\_X

- 1) CM TAA F X will be produced for each study part and for the study overall.
- 2) Sort Anatomic Class, Therapeutic Class, and Medication Terms within by descending order of overall (MRT5005 + Placebo) frequency.

```
Translate Bio, Inc.
Protocol No. MRT5005-101
```

#### Non-unique tables for CM\_TAA\_F\_X:

Table 14.3.10.2 (CM TAB F X)

Number and Percentage of Subjects with Prior Medications by Anatomic Class, Therapeutic Class, Medication Term, and Dose Group Population: Safety Analysis Set

CM F02 CM\_F03 CM F04 CM F05 CM F07 CM F08

Listing Source: CM LAA F X

#### Notes:

CM F01

- 1) CM\_TAB\_X will be produced for each study part and for the study overall.
- 2) Sort Anatomic Class, Therapeutic Class, and Medication Terms within by descending order of overall (MRT5005 + Placebo) frequency.

CFQ-R

| Part: x | | 0.0.5 | | | | 0.0.5 | | |
|---|---|---|---|---|---|---|---|---|
| | | 005 Xmg<br>N=xx | | 005 Xmg<br>=xx | | 005 Xmg<br>J=xx | | d Placebo<br>N=xx |
| | | N-AA | 11 | Absolute | 1 | V-AA | | IV-AA |
| | | Absolute | | Change | | Absolute | | Absolute |
| Visit | | Change from | | from | | Change from | | Change from |
| Statistic | Actual | Baseline | Actual | Baseline | Actual | Baseline | Actual | Baseline |
| Baseline | | | | | | | | |
| Subject 1 | XX | | XX | | XX | | XX | |
| Subject 2 | XX | | xx | | xx | | xx | |
| Subject 3 | XX | | xx | | XX | | xx | |
| Subject 4 | XX | | XX | | xx | | xx | |
| Mean | XX.X | | XX.X | | XX.X | | XX.X | |
| SD | XX.XX | | XX.XX | | XX.XX | | XX.XX | |
| Day 36 | | | | | | | | |
| Subject 1 | XX | XX | XX | XX | XX | XX | xx | XX |
| Subject 2 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 3 | XX | XX | XX | XX | XX | XX | XX | XX |
| Subject 4 | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | xx.x | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Etc. | | | | | | | | |

AB\_F06 CH\_F01 CFQ\_F01 CFQCH F01

Listing Source: QS\_LAA\_F\_X

#### Notes:

1) Include Baseline (Day -1) and Days 36, 43, 57, 85, 113, 281, and 365.

#### Footnotes

| Data<br>Type | Footnote<br>Type | Code | Prefix | Footnote |
|---|---|---|---|---|
| All | Percent | PC_F02 | Note: | Percentages were based on the number of subjects (N) in the population analyzed. |
| All | Baseline | BL_F01 | Note: | Baseline was defined as the last measurement taken prior to the first dose, obtained on or prior to the day of first dose of study drug. |
| All | Baseline | BL_F01P | Note: | Baseline was defined as the Screening measurement. |
| All | Baseline | BL_F01S | Note: | Baseline was defined as the Day -1 complete physical exam. |
| All | Change from<br>Baseline | CH_F01 | Note: | Change from baseline was defined as visit value - baseline value. |
| All | Change from<br>Baseline | CH_F02 | Note: | Relative change from baseline was defined as (visit value - baseline value)/(baseline value) $\star$ 100. |
| All | By Visit | VIS_F01 | | n = Number of subjects with the specified result at the specified visit and non-missing baseline result; nn = Number of subjects with a non-missing result at the specified visit; ( $%$ ) = Percentage of subjects with the specified result at the specified visit. |
| All | By Visit | VIS_F01a | | n = Number of subjects with the specified result at the specified visit; nn = Number of subjects with a non-missing result at the specified visit; ( $%$ ) = Percentage of subjects with the specified result at the specified visit. |
| All | Abbreviation | AB_F01 | | SD = standard deviation; SE = standard error |
| All | Abbreviation | AB_F01a | | SD = standard deviation |
| All | Abbreviation | AB_F02 | | CFTR = cystic fibrosis transmembrane conductance regulator; $FEV_1$ = forced expiratory volume in 1 second; $SD$ = standard deviation |
| All | Abbreviation | AB_F03 | | AE = adverse event; IP = investigational product; TEAE = treatment-emergent adverse event |
| All | Abbreviation | AB_F04 | | AE = adverse event; TEAE = treatment-emergent adverse event |
| All | Abbreviation | AB_F05 | | <pre>CS = clinically significant; ECG = electrocardiogram; NCS = not clinically significant</pre> |
| All | Abbreviation | AB_F06 | | <pre>CFQ-R = Cystic fibrosis questionnaire-revised; SD = standard deviation; SE = standard error</pre> |
| DS | Percent | DS_F03 | [2] | The denominator was defined as the total number of subjects who discontinued the study. |
| DM | Age | DM_F01 | [1] | Age was calculated by (date of informed consent - date of birth)/365.25, rounded down to the next largest integer using the floor function, in years. |

| Data | Footnote | | | |
|---|---|---|---|---|
| Type | Type | Code | Prefix | Footnote |
| DM | CFTR | DM_F02 | [2] | CFTR Modulator use at baseline was defined as a concomitant CFTR modulator that was in use at the start of treatment, or a CFTR modulator with missing start date. |
| CM | Percent | CM_F01 | Note: | n = Number of subjects that reported at least 1 medication within an Anatomic Class, Therapeutic Class, and Medication Term; $(\%)$ = Percentage of subjects amon the population analyzed $(N)$ . |
| CM | Count | CM_F02 | Note: | A subject that reported more than 1 medication for a particular Anatomic Class was counted only once for each Anatomic Class. |
| CM | Count | CM_F03 | Note: | A subject that reported more than 1 medication for a particular Therapeutic Class was counted only once for each Therapeutic Class. |
| CM | Count | CM_F04 | Note: | A subject that reported more than 1 medication for a particular Medication Term was counted only once for each Medication Term. |
| CM | Order | CM_F05 | Note: | Medications were presented in order of decreasing frequency, by Anatomic Class, Therapeutic Class, and Medication Term. |
| CM | Definition | CM_F06 | Note: | Concomitant medications included all medications in use at date of first study drug dose or started after date of first study drug dose, any medications that started prior to the day of first dose of study drug with missing stop date, any medications with missing start and stop dates or were classified as ongoing. |
| CM | Definition | CM_F07 | Note: | Prior medications included all medications that stopped prior to the day of first dose of the study drug, medications that started prior to the day of first dose of study drug with missing stop date or medications with missing start and stop dates. |
| CM | Dictionary | CM_F08 | Note: | Anatomic Class, Therapeutic Class, and Medication Term were based on the WHO Drug Global (2020-SEP) coding dictionary. |
| МН | Count | MH_F01 | Note: | If a subject had more than 1 medical history event within a system organ class, the subject was counted only once in that system organ class. If a subject had more than 1 medical history event that coded to the same preferred term, the subject was counted only once for that preferred term. |
| AE | Count | AE_F05 | [1] | Subjects that experienced 1 or more adverse events were counted once. |
| AE | Count | AE_F06a | [2] | If a subject experienced more than 1 adverse event, the subject was counted only once for the closest relationship to IP. AEs with missing relationships to IP were classified as being Related to IP. |
| AE | Count | AE_F06b | [3] | If a subject experienced more than 1 adverse event, the subject was counted only once for the closest relationship to nebulization/treatment administration. AEs with missing relationships were classified as being Related to nebulization/treatment administration. |

| Data<br>Type | Footnote<br>Type | Code | Prefix | Footnote |
|---|---|---|---|---|
| AE | Count | AE_F06d | [5] | If a subject experienced more than 1 adverse event classified as a pulmonary exacerbation, the subject was only counted once in the 'All' row. Subjects with both an investigator-defined and a protocol-defined TEAE classified as a pulmonary exacerbation were counted once in each row, 'Investigator-Defined' and 'Protocol-Defined'. |
| AE | Count | AE_F07 | [4] | If a subject experienced more than 1 adverse event, the subject was counted only once for the maximum severity. AEs with missing severities were counted as Severe. |
| AE | Count | AE_F07a | [2] | If a subject experienced more than 1 adverse event with a preferred term associated with the febrile reaction, the subject was counted only once for the maximum severity of any of the preferred terms contributing to the febrile reaction. AEs with missing severity were counted as Severe. |
| AE | Count | AE_F07b | [2] | If a subject experienced more than 1 hypersensitivity reaction, the subject was counted only once for the maximum severity of any of the hypersensitivity reactions. AEs with missing severity were counted as Severe. |
| AE | Order | AE_F08 | Note: | Incidences were displayed in descending order of frequency of System Organ Class and by Preferred Term within System Organ Class. |
| AE | Order | AE_F09 | Note: | Incidences were displayed in descending order of frequency of Preferred Term. |
| AE | Dictionary | AE_F14 | Note: | System Organ Class and Preferred Term were based on the Version 23.1 of the MedDRA coding dictionary. |
| AE | Dictionary | AE_F14a | Note: | Preferred Term was based on the Version 23.1 of the MedDRA coding dictionary. |
| AE | Interval | AE_F15 | Note: | Time intervals were determined by the start day of the adverse event. |
| AE | Count | AE_F16 | Note: | n represents the number of subjects that experienced an adverse event in a given category. m represents the number of adverse events in a given category. |
| AE | Definition | AE_F17a | Note: | Febrile reactions were identified based on a preferred term of body temperature increased or preferred term of pyrexia within the 24 hours after completion of nebulization on any dosing day with at least one other systemic symptom reported as a preferred term of headache, arthralgia, myalgia, fatigue, chills, nausea, or vomiting within the 24 hours after completion of nebulization on any dosing day. |
| AE | Definition | AE_F17b | Note: | Hypersensitivity reactions were identified based on a preferred term of hypersensitivity within the 24 hours after completion of nebulization on any dosing day. |
| AE | Definition | AE_F17c | [2] | Severity grade for each febrile reaction was based on the maximum severity of the preferred terms comprising the febrile reaction. Febrile reactions with missing severity were counted as Severe. |

| Data | Footnote | | | |
|---|---|---|---|---|
| Type | Type | Code | Prefix | Footnote |
| AE | Interval | AE_F18 | Note: | The 1 month post-dose time interval is defined as through Day 29 for Part A, through Day 57 for Part B, through Day 32 for Part D. |
| AE | Count | AE_F19 | Note: | N represents the number of subjects in a given dose group that experienced an adverse event. |
| EG | Baseline | EG_F01 | Note: | The baseline value was defined as the Day -1 ECG measurement. |
| EG | Baseline | EG_F01D | Note: | The baseline value was defined as the screening ECG measurement. |
| EG | Schedule | EG_F02 | Note: | Only ECGs scheduled per the protocol were summarized. |
| EX | Count | EX_F01 | Note: | Full dose refers to completion of all nebulizers as planned; partial dose refers to incomplete nebulization. Full and partial dose are independent of the presence or absence of excess residual in the medication chamber. |
| VS | Schedule | VS_F01 | Note: | The final recording during nebulization for blood pressure, pulse rate, and pulse oximetry was counted as the 'DAY 1 (0 HR POST-DOSE)' value. |
| RE | Baseline | RE_F01 | [1], [3] | The baseline value was defined as the average of the results from testing on Day - ${\bf 1}$ and at pre-dose on Day 1. |
| RE | Baseline | RE_F01D | [1],[3] | The baseline value was defined as the result from testing pre-dose on Day 1. |
| RE | Baseline | RE_F010 | [1],[3] | The baseline value was defined as the average of the results from testing on Day - 1 and at pre-dose on Day 1 for Part A and Part B, and defined as the result from testing pre-dose on Day 1 for Part D. |
| CFQ | Baseline | CFQ_F01 | Note: | The baseline value was defined as the Day -1 CFQ-R respiratory domain score. |
| CFQ | Baseline | CFQCH_F01 | Note: | At baseline, all subjects with baseline data contributed to the reported baseline mean. For each visit, the mean actual value was the mean across all subjects with data at that visit. The change from baseline was calculated for each subject with data at baseline and that visit, then reported as a mean change. |
| XR | Schedule | XR_F01 | Note: | Only chest x-rays scheduled per the protocol were summarized. |

# Translate Bio, Inc. PROTOCOL NUMBER MRT5005-101

A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled, Combined Single and Multiple Ascending Dose Study Evaluating the Safety, Tolerability, and Biological Activity of MRT5005 (mRNA/mr LNP) Administered by Nebulization to Adult with ic Fibrosis

### Listing Specifications

VERSION DATE: 26 October 2021

SPONSOR: Translate Bio, Inc. 29 Hartwell Avenue Lexington, MA 02421 Telephone: (617) 945-7361

PREPARED BY: Rho, Inc. 2635 E NC Hwy 54 Durham, NC 27713 Telephone: (919) 408-8000 Fax: (919) 408-0999

### Listing Specifications

#### Table of Contents

| General Programming Notes | 3 |
|---|---|
| Listing 16.2.1.1 (DS LAA F X) Listing of Screen Failures | |
| Listing 16.2.1.2 (DS LAB F X) Listing of Subject Disposition | 5 |
| Listing 16.2.1.3 (DS LAC F X) Listing of Visits Not Done, Conducted as Home Health Visits, or Visits Conducted as Telephone Vis | |
| as a Replacement for a Scheduled In-Clinic Visit | 6 |
| Listing 16.2.2 (PD LAA F X) Listing of Protocol Deviations | 7 |
| Listing 16.2.4.1 (DM LAB F X) Listing of Demographics and Baseline Characteristics | 8 |
| Listing 16.2.5.1 (EX_LAB_F_B, EX_LAB_F_D) Listing of Overall Extent of Exposure | |
| Listing 16.2.5.2 (EX_LAC_F_X) Listing of Extent of Exposure at the Visit Level | 10 |
| Listing 16.2.5.3 (EX_LAA F X) Listing of Investigational Product Administration | 11 |
| Listing 16.2.6.1 (MH LAA F X) Listing of Medical History by Subject, System Organ Class, and Preferred Term | 12 |
| Listing 16.2.7.1 (AE LAA F X) Listing of Adverse Events by Subject, System Organ Class, and Preferred Term | 13 |
| Listing 16.2.7.2 (AE LAB F X) Listing of Adverse Events Leading to Treatment Discontinuation by Subject, System Organ Class, an | nd |
| Preferred Term | |
| Listing 16.2.7.3 (AE LAD F X) Listing of Adverse Events Resulting in Death by Subject, System Organ Class, and Preferred Term. | 14 |
| Listing 16.2.7.4 (AE LAC F X) Listing of Serious Adverse Events by Subject, System Organ Class, and Preferred Term | 14 |
| Listing 16.2.7.5 (AE LAL F X) Listing of Adverse Events of Special Interest by Subject, System Organ Class, and Preferred Term . | 14 |
| Listing 16.2.7.6 (AE LAF F X) Listing of Adverse Events Classified as Pulmonary Exacerbations (Investigator and Protocol-Define | ed) |
| by Subject, System Organ Class, and Preferred Termby Subject, System Organ Class, and Preferred Term | 14 |
| Listing 16.2.7.7 (AE_LAI_F_X) Listing of Pyrexia or Elevated Body Temperature Adverse Events Reported During and Up To 24 Hours | s |
| After Completion of Nebulization by Subject, System Organ Class, and Preferred Term | |
| Listing 16.2.7.8 (AE_LAJ_F_X) Listing of Adverse Events Reported During and Up To 24 Hours After Completion of Nebulization by | |
| Subject, System Organ Class, and Preferred Term | |
| Listing 16.2.7.9 (AE_LAK_F_X) Listing of Febrile Reactions and Hypersensitivity Reactions in First 24 Hours After Completion of | |
| Nebulization by Subject and Preferred Term | |
| Listing 16.2.8.1 (LB_LAA_F_X) Listing of Chemistry Values | |
| Listing 16.2.8.2 (LB_LAB_F_X) Listing of Hematology Values | |
| Listing 16.2.8.3 (LB_LAC_F_X) Listing of Urinalysis Values | |
| Listing 16.2.8.4 (LB_LAD_F_B, LB_LAD_F_D) Listing of Coagulation Values | |
| Listing 16.2.8.5 (LB_LAE_F_B, LB_LAE_F_D) Listing of Serum Inflammatory Markers | |
| Listing 16.2.8.8 (PG_LAA_F_X) Listing of Pregnancy Results | |
| Listing 16.2.9.1 (VS_LAA_F_X) Listing of Vital Signs | |
| Listing 16.2.10.1 (EG_LAA_F_X) Listing of Overall Electrocardiogram Interpretation Findings | |
| Listing 16.2.11.1 (CX_LAA_F_X) Listing of Chest X-Ray Findings | |
| Listing 16.2.12.1 (PE_LAA_F_X) Listing of Physical Examination Results | |
| Listing 16.2.13.1 (RE_LAA_F_X) Listing of Spirometry Values | |
| Listing 16.2.14.1 (CM_LAA_F_X) Listing of Prior and Concomitant Medications | |
| Listing 16.2.14.2 (CM_LAB_F_X) Listing of Concomitant Surgical Procedures | |
| Listing 16 2 15 1 (OS LAA F R) Listing of CFO-R Respiratory Domain Scores | 29 |

#### General Programming Notes

The following instructions apply to all listing displays.

#### DISPLAY OUTPUTS FOR EACH PART

Each listing will be produced for each study part (A, B, D), unless otherwise specified. Listings will not be produced for the study overall. Each version of the listing will include the relevant study part in the header and in the listing identifier. For example, DS\_LAA\_F\_X will be identified as DS\_LAA\_F\_A for Part A and will include a header to show 'Part A'. A, B or D will be added to each display number.

#### PROGRAMMER NOTES

Programmer notes appear at the bottom of each listing display shell where applicable.

Dose groups for each part are as follow:

- Part A: MRT5005 8mg, MRT5005 16mg, MRT5005 20mg, MRT5005 24mg, Pooled Placebo
- Part B: MRT5005 8mg, MRT5005 12mg, MRT5005 16mg, MRT5005 20mg, Pooled Placebo
- Part D: MRT5005 4mg, Placebo

The maximum number of decimal places reported will be 4.

#### PAGE FORMATTING

The specifications for the format of each page are page size=47, line size=134, font=Courier, font size=8, and margin = 1.5" top, 1" bottom, left, and right.

"Dataset Source: <Dataset Name>" will be printed on the right side of the footer for each listing.

#### SORTING

Unless otherwise specified, listings are sorted by Subject Number, Visit Number, in that order when the variables are included in the table. Only show the value of a sort-variable when it changes or when a new page starts. Insert a blank row between the data for subjects.

#### Listing 16.2.1.1 (DS\_LAA\_F\_X) Listing of Screen Failures Population: Screened Subjects

Part: x

| Subject Number | Date of Informed<br>Consent | Date of Screen<br>Failure | Reason for Screen<br>Failure/Other, Specify |
|---|---|---|---|
| xxxx | YYYY-MM-DD | YYYY-MM-DD | XXXXXXX/XXXXX |
| XXXX | YYYY-MM-DD | YYYY-MM-DD | XXXXXXX/XXXXX |
| Etc. | | | |

Dataset Source: ADSL

Listing 16.2.1.2 (DS\_LAB\_F\_X)
Listing of Subject Disposition
Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Date of<br>Informed<br>Consent | Date of Randomization/ Date of First Dose of Study Drug | Date of Last<br>Dose of Study<br>Drug/<br>Study Day [1] | Did<br>subject<br>receive<br>all study<br>treatment? | Date of<br>Completion or<br>Early<br>Termination/<br>Study Day [2] | Completed the study? | Reason for Study<br>Withdrawal/Other,<br>Specify |
|---|---|---|---|---|---|---|---|
| XXXX | YYYY-MM-<br>DD | YYYY-MM-DD/<br>YYYY-MM-DD | YYYY-MM-DD/<br>XX | Yes | YYYY-MM-DD/<br>XX | Yes | XXXXXXX/<br>XXXXX |
| xxxx | YYYY-MM-<br>DD | YYYY-MM-DD/<br>YYYY-MM-DD | YYYY-MM-DD/<br>XX | No | YYYY-MM-DD/<br>XX | No | XXXXXXX/<br>XXXXXXXX |

Etc.

[1] DS\_L01 [2] DS\_L02

Dataset Source: ADSL

#### Notes:

1) Dose groups are specified in the general programming notes.

#### Listing 16.2.1.3 (DS\_LAC\_F\_X)

Listing of Visits Not Done, Conducted as Home Health Visits, or Visits Conducted as Telephone Visits as a Replacement for a Scheduled In-Clinic Visit

Population: Safety Analysis Set

Part: x
Dose Group: xxx

| | | | Visit Not Done | |
|----------------|----------|------------|----------------|--------------|
| Subject Number | Visit | Visit Date | or Visit Type | Reason |
| XXXX | XXXXXXXX | YYYY-MM-DD | XXXXXX | XXXXXXXXXXXX |
| | | | | xxxxxxxxxxxx |
| XXXX | XXXXXXXX | YYYY-MM-DD | XXXXXX | xxxxxxxxxxxx |
| | | | | XXXXXXXXXXXX |
| Etc. | | | | |

Dataset Source: VE, SUPPVE

- 1) Dose groups are specified in the general programming notes.
- 2) List any visits not done, conducted as home health visit, or visit conducted as a telephone visit as a replacement for a scheduled in-clinic visit.

Listing 16.2.2 (PD\_LAA\_F\_X) Listing of Protocol Deviations Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Date<br>Deviation<br>was<br>Discovered | Associated Study Visit/ Date Deviation Started | Protocol Deviation Type/ Protocol Deviation Description | Corrective/Preventative<br>Action | Reportable to the IRB?/<br>Date IRB Notified |
|---|---|---|---|---|---|
| XXXX | YYYY-MM-DD | XXXXXX/<br>YYYY-MM-DD | XXXXXXXXXXXXX/<br>XXXXXXXXXXXXX | XXXXXXXXXXXX | No/ |
| XXXX | YYYY-MM-DD | XXXXXX/<br>YYYY-MM-DD | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX | xxxxxxxxxxxx | Yes/<br>YYYY-MM-DD |
| Etc. | | | | | |

Dataset Source: DV, SUPPDV

- 1) Dose groups are specified in the general programming notes.
- 2) Listing will include both blinded and unblinded protocol deviations

# Listing 16.2.4.1 (DM\_LAB\_F\_X) Listing of Demographics and Baseline Characteristics Population: Safety Analysis Set

Part: x

Dose Group: xx

| | | | | | | | | Genotype | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Date of<br>Randomization | Date<br>of<br>Birth | Age<br>[1] | Sex | Race/<br>Ethnicity | CFTR Modulator<br>Use | Baseline<br>Percent<br>Predicted FEV <sub>1</sub><br>[2] | First Mutation<br>Class/Second<br>Mutation Class | First Mutation<br>Name/Second<br>Mutation Name |
| XXXX | YYYY-MM-DD | YYYY-<br>MM-DD | XX | Male | White/<br>Hispanic or<br>Latino | Yes | XX.X | XXX/XXX | XXX/XXX |
| XXXX | YYYY-MM-DD | YYYY-<br>MM-DD | XX | Female | Other:<br>XXXXXXXXXX/<br>Not<br>Hispanic or<br>Latino | No | XX.X | xxx/xxx | XXX/XXX |

Etc.

DM L02

[1] DM\_L01

[2] RE L02

Dataset Source: ADSL

#### Notes:

1) Dose groups are specified in the general programming notes.

# Listing 16.2.5.1 (EX\_LAB\_F\_B, EX\_LAB\_F\_D) Listing of Overall Extent of Exposure Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Number of Full Doses<br>Administered | Number of Partial Doses<br>Administered |
|---|---|---|
| XXXX | XX | XX |
| XXXX | XX | XX |
| Etc. | | |

Note: EX F01

Dataset Source: ADEXSUM

#### Notes:

1) Dose groups are specified in the general programming notes.

# Listing 16.2.5.2 (EX\_LAC\_F\_X) Listing of Extent of Exposure at the Visit Level Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Date of IP<br>Administration | Was Full Dose | Reason Full Dose Was | Actual Number of Medication<br>Chambers Completed/<br>Expected Number of<br>Medication Chambers |
|---|---|---|---|---|---|
| Subject Number | Visit | /Study Day | Administered? | Not Administered | Completed |
| XXXX | | YYYY-MM-DD/<br>XX | Yes | | xx/xx |
| XXXX | | YYYY-MM-DD/<br>XX | No | xxxxxx | xx |
| XXXX | | YYYY-MM-DD/<br>XX | Yes | | xx |

Etc.

Note: EX\_L01 Note: EX\_L02 Note: EX\_F01

Dataset Source: ADEXVIS
## Listing 16.2.5.3 (EX\_LAA\_F\_X) Listing of Investigational Product Administration Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Visit | Start<br>Date/Time of<br>Nebulizer/<br>Study Day | End Date/Time<br>of Nebulizer/<br>Study Day | Nebulization<br>Complete | Excess Residual in Medication Chamber? |
|---|---|---|---|---|---|
| XXXX | | YYYY-MM-DD/<br>XX | YYYY-MM-DD/<br>XX | Yes | No |
| | | YYYY-MM-DD/<br>XX | YYYY-MM-DD/<br>XX | Yes | No |
| | | YYYY-MM-DD/<br>XX | YYYY-MM-DD/<br>XX | No | Yes |
| XXXX | | YYYY-MM-DD/<br>XX | YYYY-MM-DD/<br>XX | Yes | No |

Etc

Note: EX F01

Dataset Source: ADEX

- 1) Dose groups are specified in the general programming notes.
- 2) Remove fully missing records.

### 

Part: x

Dose Group: xxx

| Subject Number | System Organ<br>Class/<br>Preferred Term | Medical History<br>Event | Start<br>Date/<br>Study Day | End<br>Date/<br>Study<br>Day | Ongoing? |
|---|---|---|---|---|---|
| XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | YYYY-MM-<br>DD/<br>XX | YYYY-MM-<br>DD/<br>XX | No |
| XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXX | YYYY-MM-<br>DD/<br>XX | | Yes |
| ELC. | | | | | |

Note: AE L03

Dataset Source: ADMH

- 1.) Sort by Dose Group, Subject Number, Start Date, Stop Date, System Organ Class, Preferred Term.
- 2.) Dose groups are specified in the general programming notes.

## Listing 16.2.7.1 (AE\_LAA\_F\_X) Listing of Adverse Events by Subject, System Organ Class, and Preferred Term Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Start Date/Start Time/Study Day End Date/ End Time/ Study Day/ Ongoing? | System Organ<br>Class/<br>Preferred<br>Term/<br>Verbatim<br>Term | AE<br>Duration<br>(days) | Severity/<br>Action<br>Taken | Outcome/<br>Specify | Relation<br>ship to<br>IP | Relationship to<br>Nebulization/<br>Treatment<br>Administration | Serious<br>AE? | Treatment-<br>Emergent? |
|---|---|---|---|---|---|---|---|---|---|
| XXXX | YYYY-MM- DD/HH:MM:SS / XX/ YYYY-MM-DD/ HH:MM:SS/XX / No | XXXXXXXXXXX<br>XXX/<br>XXXXXXXXXXX<br>XXX/<br>XXXXXX | XX | xxxxxx/<br>xxxxxxx | XXXXXX/ | XXXXXXXX<br>X | xxxxxxxx | Yes | Yes |
| XXXX | YYYY-MM-DD/<br>HH:MM:SS/XX<br>/<br>YYYY-MM-DD/<br>HH:MM:SS/XX<br>/<br>No | XXXXXXXXXXX<br>XXX/<br>XXXXXXXXXXXX<br>XXX/<br>XXXXXX | XX | xxxxxx/<br>xxxxxx | XXXXXX/<br>XXXX | XXXXXXXX | xxxxxxxx | No | No |
| Etc. | | | | | | | | | |

Note: AE\_L01 Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

- 1.) Sort by Dose Group, Subject Number, Start Date, Stop Date, System Organ Class, Preferred Term, Verbatim Term.
- 2.) Dose groups are specified in the general programming notes.

#### Non-unique listings for (for AE\_LAA):

Listing 16.2.7.2 (AE LAB F X)

Listing of Adverse Events Leading to Treatment Discontinuation by Subject, System Organ Class, and Preferred Term

Population: Safety Analysis Set

Note: AE\_L01 Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

Listing 16.2.7.3 (AE LAD F X)

Listing of Adverse Events Resulting in Death by Subject, System Organ Class, and Preferred Term

Population: Safety Analysis Set

Note: AE\_L01 Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

Listing 16.2.7.4 (AE LAC F X)

Listing of Serious Adverse Events by Subject, System Organ Class, and Preferred Term

Population: Safety Analysis Set

Note: AE\_L01 Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

Listing 16.2.7.5 (AE\_LAL\_F\_X)

Listing of Adverse Events of Special Interest by Subject, System Organ Class, and Preferred Term

Population: Safety Analysis Set

Note: AE\_L01 Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

Listing 16.2.7.6 (AE LAF F X)

Listing of Adverse Events Classified as Pulmonary Exacerbations (Investigator and Protocol-Defined) by Subject, System Organ Class,

and Preferred Term

Population: Safety Analysis Set

Note: AE\_L01

Note: AE\_L02 Note: AE\_L03

Dataset Source: ADAE

#### Notes:

1.) Add "Type" to the Treatment Emergent column with values of "Investigator-Defined" and "Protocol-Defined".

#### Listing 16.2.7.7 (AE LAI F X)

Listing of Pyrexia or Elevated Body Temperature Adverse Events Reported During and Up To 24 Hours After Completion of Nebulization by Subject, System Organ Class, and Preferred Term

Population: Safety Analysis Set

## Part: x Dose Group: xxx

| Subject Number | Start Date/Start Time/Study Day End Date/ End Time/ Study Day/ Ongoing? | Start Time<br>Relative to<br>End of<br>Nebulization<br>(Hours) [1] | System Organ<br>Class/<br>Preferred<br>Term/<br>Verbatim<br>Term | Severity/<br>Action<br>Taken | Outcome/<br>Specify | Relation<br>ship to<br>IP | Relationship to<br>Nebulization/<br>Treatment<br>Administration | Serious<br>AE? |
|---|---|---|---|---|---|---|---|---|
| XXXX | YYYY-MM- DD/HH:MM:SS / XX/ YYYY-MM-DD/ HH:MM:SS/XX / No | XX | XXXXXXXXXXX<br>XXX/<br>XXXXXXXXXX/<br>XXXXXXXXXX | xxxxxx/<br>xxxxxx | XXXXXX/ | XXXXXXXX<br>X | xxxxxxxx | Yes |
| xxxx | YYYY-MM-DD/<br>HH:MM:SS/XX<br>/<br>YYYY-MM-DD/<br>HH:MM:SS/XX<br>/<br>No | <br>N/A (During) | XXXXXXXXXXXX XXX XXXXXXXXXX/ XXXXXXXX | xxxxxx/<br>xxxxxx | XXXXXX/<br>XXXX | xxxxxxxx | xxxxxxxx | No |
| Etc. | | | | | | | | |

[1] AE\_L06
Note: AE\_L01
Note: AE\_L03
Note: AE\_L04

Dataset Source: ADAE

- 1.) Sort by Dose Group, Subject Number, Start Date, Stop Date, System Organ Class, Preferred Term, Verbatim Term.
- 2.) Dose groups are specified in the general programming notes.

- 3.) For any subject with an AE of Pyrexia or Elevated Body Temperature within 24 hours after dosing, include all other AEs for that subject that occurred within 24 hours after dosing.
- 4.) Add footnote reference [1] to column 3.
- 5.) Round start time relative to end of nebulization (hours) to 2 decimal places.

Listing 16.2.7.8 (AE LAJ F X)

Listing of Adverse Events Reported During and Up To 24 Hours After Completion of Nebulization by Subject, System Organ Class, and

Preferred Term

Population: Safety Analysis Set

[1] AE\_L06 Note: AE\_L01 Note: AE\_L03

Dataset Source: ADAE

#### Notes:

- 1.) Sort by Dose Group, Subject Number, Start Date, Stop Date, System Organ Class, Preferred Term, Verbatim Term.
- 2.) Dose groups are specified in the general programming notes.
- 3.) Include any AE that occurred during nebulization or within 24 hours after dosing.
- 4.) Add footnote reference [1] to column 3.
- 5.) Round start time relative to end of nebulization (hours) to 2 decimal places.

Listing 16.2.7.9 (AE LAK F X)

Listing of Febrile Reactions and Hypersensitivity Reactions in First 24 Hours After Completion of Nebulization by Subject and Preferred Term

Population: Safety Analysis Set

[1] AE\_L08 Note: AE\_L01 Note: AE\_L03

Dataset Source: ADAE

- 1.) Sort by Dose Group, Subject Number, Start Date, Stop Date, System Organ Class, Preferred Term, Verbatim Term.
- 2.) Dose groups are specified in the general programming notes.
- 3.) For any subject with a febrile reaction or hypersensitivity reaction during or within 24 hours after dosing, include all other AEs that meet the criteria for febrile reaction or hypersensitivity reaction for that subject that occurred during nebulization or within 24 hours after dosing.
- 4.) Add footnote reference [1] to column 3.

## Listing 16.2.8.1 (LB\_LAA\_F\_X) Listing of Chemistry Values Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject Number | Visit | Date/Time of<br>Assessment/<br>Study Day | Lab Test<br>(units) | Result | Classification/<br>CS?/<br>Comment | Reference Range |
|---|---|---|---|---|---|---|
| XXXX | | YYYY-MM-<br>DD/HH:MM:SS | Albumin | XXX | | |
| | | | Alkaline<br>Phosphatase | XXX | | |
| | | | ALT | XXX | | |
| | | | AST | XXX | | |
| | | | Blood Urea<br>Nitrogen | XXX | | |
| | | YYYY-MM-<br>DD/HH:MM:SS | | XXX | | |
| | | YYYY-MM-<br>DD/HH:MM:SS | | XXX | | |
| XXXX | | YYYY-MM-<br>DD/HH:MM:SS | | XXX | | |

Etc.

CS\_01 Note: LB 01

Dataset Source: ADLB

- 1) Laboratory parameters are listed alphabetically.
- 2) Dose groups are specified in the general programming notes.

#### Non-unique listings for LB\_LAA:

Listing 16.2.8.2 (LB\_LAB\_F\_X) Listing of Hematology Values Population: Safety Analysis Set

CS\_01 Note: LB\_01

Dataset Source: ADLB

Listing 16.2.8.3 (LB\_LAC\_F\_X) Listing of Urinalysis Values Population: Safety Analysis Set

CS\_01 Note: LB\_01

Dataset Source: ADLB

Listing 16.2.8.4 (LB\_LAD\_F\_B, LB\_LAD\_F\_D)
Listing of Coagulation Values
Population: Safety Analysis Set

CS\_01 Note: LB 01

Dataset Source: ADLB

## Listing 16.2.8.5 (LB\_LAE\_F\_B, LB\_LAE\_F\_D) Listing of Serum Inflammatory Markers Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Date/Time of Assessment/ | Marker | Result | Reference |
|---|---|---|---|---|---|
| Subject Number | Visit | Study Day | | | Range |
| XXXX | | YYYY-MM-DD/HH:MM:SS | Interferon | XXX | |
| | | | Interleukin-1B | XXX | |
| | | | Interleukin-2 | XXX | |
| | | | Interleukin-4 | XXX | |
| | | | Interleukin-6 | XXX | |
| | | | Interleukin-8 | XXX | |
| | | | Interleukin-10 | XXX | |
| | | | Interleukin-12p70 | XXX | |
| | | | Interleukin-13 | XXX | |
| | | | Tumor Necrosis Factor | XXX | |
| | | YYYY-MM-DD/HH:MM:SS | | XXX | |
| | | YYYY-MM-DD/HH:MM:SS | | XXX | |
| XXXX | | YYYY-MM-DD/HH:MM:SS | | XXX | |
| Etc. | | | | | |

Dataset Source: ADLB

- 1) Inflammatory markers are listed alphabetically.
- 2) Dose groups are specified in the general programming notes.

Listing 16.2.8.8 (PG\_LAA\_F\_X)
Listing of Pregnancy Results
Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Date of Assessment/ | Was the Pregnancy | Pregnancy Test |
|---|---|---|---|---|
| Subject Number | Visit | Study Day | Test Completed? | Result |
| XXXX | | YYYY-MM-DD/XX | Yes | Negative |
| | | YYYY-MM-DD/XX | Yes | Negative |
| XXXX | | YYYY-MM-DD/XX | Yes | Negative |
| Etc. | | | | |

Dataset Source: ADLB

## Listing 16.2.9.1 (VS\_LAA\_F\_X) Listing of Vital Signs Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject | Visit/ | Visit<br>Date/Time/ | Systolic Blood<br>Pressure<br>(mmHg)/<br>Diastolic<br>Blood Pressure | Pulse<br>Rate | Respiratory<br>Rate | Temperature | Pulse<br>Oximetry | Weight |
|---|---|---|---|---|---|---|---|---|
| Number | Timepoint | Study Day | (mmHg) | (bpm) | (breaths/min) | (C) | (왕) | (kg) |
| XXXX | | YYYY-MM- DD/HH:MM:SS | | | | | | |
| XXXX | | YYYY-MM- DD/HH:MM:SS | | | | | | |
| Etc. | | | | | | | | |

Dataset Source: ADVS

## 

Part: x
Dose Group: xxx

| se Gloup, xxx | | | |
|----------------|-------|-------------|--------|
| | | Date of | |
| | | Assessment/ | |
| Subject Number | Visit | Study Day | Result |
| XXXX | | YYYY-MM-DD/ | |
| | | XX | |
| | | YYYY-MM-DD/ | |
| | | XX | |
| | | YYYY-MM-DD/ | |
| | | XX | |
| XXXX | | YYYY-MM-DD/ | |
| | | XX | |
| Etc. | | | |

CS\_01

Dataset Source: ADEG

Listing 16.2.11.1 (CX\_LAA\_F\_X)
Listing of Chest X-Ray Findings
Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Date of | | |
|----------------|-------|-------------|--------|---------|
| | | Assessment/ | | Details |
| Subject Number | Visit | Study Day | Result | |
| XXXX | | YYYY-MM-DD/ | | |
| | | XX | | |
| | | YYYY-MM-DD/ | | |
| | | XX | | |
| | | YYYY-MM-DD/ | | |
| | | XX | | |
| XXXX | | YYYY-MM-DD/ | | |
| | | XX | | |
| Etc. | | | | |

CS\_01

Dataset Source: ADCX

## Listing 16.2.12.1 (PE\_LAA\_F\_X) Listing of Physical Examination Results Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Date of | | | |
|----------------|-------|--------------|-------------|---------|-------------|
| | | Assessment/ | Body System | | |
| Subject Number | Visit | Study Day | Examined | Result | Description |
| XXX | | YYYY-MM-DD/ | General | | |
| | | XX | Appearance | XXXXXX | xxxxxx |
| | | | Skin | XXXXXXX | xxxxxx |
| | | | Etc. | | |
| | | WWW 104 DD / | | | |
| | | YYYY-MM-DD/ | | | |
| | | XX | | | |
| XXXX | | YYYY-MM-DD/ | | | |
| | | XX | | | |
| | | 2121 | | | |
| E+ a | | | | | |
| Etc. | | | | | |

\_\_

CS\_01 PE L01

Dataset Source: ADPE

Listing 16.2.13.1 (RE\_LAA\_F\_X) Listing of Spirometry Values Population: Safety Analysis Set

Part: x
Dose Group: xxx

| Subject Number | Visit | Date/Time of<br>Assessment/<br>Study Day | Spirometry<br>Test [1] | Result | Reference<br>Result |
|---|---|---|---|---|---|
| xxxx | | YYYY-MM-<br>DD/HH:MM:SS/ | FEF2575 | XXX | |
| | | XX | FET | XXX | |
| | | | FEV1 | XXX | |
| | | | FEV1FVC | | |
| | | YYYY-MM-<br>DD/HH:MM:SS/<br>XX | | XXX | |
| | | YYYY-MM-<br>DD/HH:MM:SS/<br>XX | | XXX | |
| XXXX | | YYYY-MM-<br>DD/HH:MM:SS/<br>XX | | XXX | |
| Etc. | | | | | |

[1] RE\_L01 Note: RE\_L02 Note: RE\_L03

Dataset Source: ADRE

- 1) For RE\_LAA\_D, remove footnote RE\_LO2.
- 2) Present Baseline-Derived after Day 1 (pre-dose)

## Listing 16.2.14.1 (CM\_LAA\_ $F_X$ ) Listing of Prior and Concomitant Medications Population: Safety Analysis Set

Part: x

Dose Group: xxx

| | | Start | | | | | |
|---|---|---|---|---|---|---|---|
| | | Date (Study | | | | | |
| | | Day)/ | | | | | |
| | Anatomic Class/ | Stop Date | | Dose/ | | | |
| | Therapeutic Class/ | (Study | | Unit/ | | | |
| Subject | Preferred Name/ | Day) / | Prior or | Dose | | Route/ | Taken for |
| Number | Verbatim Term | Ongoing? | Concomitant? | Form | Indication | Frequency | AE? |
| XXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM- | Concomitant | XXX/ | XXXXXXXX | XXXXXXXXX/ | Yes |
| | XXXXXXXXXXXXXXXXXXXXXXX/ | DD/ | | XXX/ | | XXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXX/ | Yes | | XXX | | | |
| | XXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM- | Prior | XXX/ | XXXXXXXX | XXXXXXXXX/ | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX/ | DD/ | | XXX/ | | XXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX/ | YYYY-MM-DD | | XXX | | | |
| | XXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| XXXX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx/ | YYYY-MM- | Concomitant | XXX/ | XXXXXXXXX | XXXXXXXXX/ | No |
| | XXXXXXXXXXXXXXXXXXXXXXX/ | DD/ | | XXX/ | | XXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXX/ | YYYY-MM-DD | | XXX | | | |
| | XXXXXXXXXXXXXXXXXXXXXXX | | | | | | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD | Concomitant | XXX/ | XXXXXXXX | XXXXXXXXX/ | No |
| | XXXXXXXXXXXXXXXXXXXXXXXXXX/ | | | XXX/ | | XXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXX/ | | | XXX | | | |
| | XXXXXXXXXXXXXXXXXXXXXX | | | | | | |

Note: CM\_L01 Note: CM\_L02

Dataset Source: ADCM

## Listing 16.2.14.2 (CM LAB\_F\_X) Listing of Concomitant Surgical Procedures Population: Safety Analysis Set

Part: x

Dose Group: xxx

| Subject<br>Number | System Organ Class/<br>Preferred Term/<br>Procedure | Start Date (Study Day)/<br>Stop Date (Study Day) | Indication |
|---|---|---|---|
| XXXX | xxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxxxx/<br>xxxxxx | YYYY-MM-DD (XX)/<br>YYYY-MM-DD (XX) | xxxxxxxx |
| | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXX | YYYY-MM-DD (XX)/<br>YYYY-MM-DD (XX) | xxxxxxxx |
| XXXX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXX/<br>XXXXXX | YYYY-MM-DD (XX)/<br>YYYY-MM-DD (XX) | xxxxxxxx |

Note: AE L03

Dataset Source: PR

## Listing 16.2.15.1 (QS\_LAA\_F\_B) Listing of CFQ-R Respiratory Domain Scores Population: Safety Analysis Set

Part: x

| Subject | | Date of Assessmen | t/ | |
|---|---|---|---|---|
| Number | Visit | Study Day | Question | Response |
| XXXX | XXXXXXX | YYYY-MM-DD/<br>XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX |
| | | | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX |
| | | | Respiratory Domain Score | XXX |
| XXXX | XXXXXXX | YYYY-MM-DD/<br>XX | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | XXX |
| | | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXX |
| | | | Respiratory Domain Score | XXX |

QS F01

Dataset Source: ADQS

- 1) Include questions that contribute to the respiratory domain score.
- 2) Include all visits (Baseline and Days 36, 43, 57, 85, 113, 197, 281, 365).

#### Footnotes

| Data<br>Type | Footnote Type | Code | Prefix | Footnote |
|---|---|---|---|---|
| DS | Study day | DS_L01 | [1] | Study day of last dose of study drug was defined as treatment end date - treatment start date + 1. |
| DS | Study day | DS_L02 | [2] | Study day was defined as date of completion or early termination - treatment start date $+\ 1$ . |
| DM | Derivation | DM_L01 | [1] | Age is calculated by (date of informed consent - date of birth)/365.25, rounded down to the next largest integer using the floor function, in years. |
| DM | Abbreviation | DM_L02 | | CFTR = cystic fibrosis transmembrane conductance regulator. |
| EX | Schedule | EX_L01 | Note: | For the 4 mg dose group, 1 medication chamber was expected. For the 8 mg dose group, 2 medication chambers were expected. For the 12 mg dose group, 3 medication chambers were expected. For the 16 mg dose group, 4 medication chambers were expected. For the 20 mg dose group, 5 medication chambers were expected. For the 24 mg dose group, 6 medication chambers were expected. |
| EX | Derivation | EX_L02 | Note: | A medication chamber was counted as completed if nebulization was marked as completed and there was no excess residual in the medication chamber. The medication chamber is the cup recorded on the investigational product administration case report form page. |
| EX | Count | EX_F01 | Note: | Full dose refers to completion of all nebulizers as planned; partial dose refers to incomplete nebulization. Full and partial dose are independent of the presence or absence of excess residual in the medication chamber. |
| AE | Study day | AE_L01 | Note: | Start day and end day of AEs were defined relative to the date of first dose of study drug. |
| AE | Derivation | AE_L02 | Note: | AE Duration (days) was calculated as AE end date - AE start date + 1. Imputed AE start dates and imputed AE end dates were used in the case of partially missing dates. Any duration calculation that required use of imputed AE start date or imputed AE end date were identified by `*'. |
| AE | Dictionary | AE_L03 | Note: | System Organ Class and Preferred Term are based on the Version 23.1 of the MedDRA coding dictionary. |
| AE | Definition | AE_L04 | Note: | All adverse events that occurred within the 24 hours after completion of nebulization for subjects that had an adverse event of pyrexia within the 24 hours after completion of nebulization are listed. |
| AE | Definition | AE_L06 | [1] | 'N/A (During)' indicates that the adverse event occurred during nebulization. |
| AE | Definition | AE_L08 | [1] | All adverse events that met the criteria for a febrile reaction or hypersensitivity reaction that occurred within the 24 hours after completion of |

| Data | Footnote Type | | | |
|---|---|---|---|---|
| Type | | Code | Prefix | Footnote |
| | | | | nebulization for subjects that had a febrile reaction or hypersensitivity reaction within the 24 hours after completion of nebulization are listed. |
| LB, CS | Abbreviation | CS_01 | | CS = clinically significant; NCS = not clinically significant |
| LB | Definition | LB_01 | Note | The classification of Low, Normal, or High was based on the global laboratory reference ranges used across all sites. Clinical significance was assessed for out of range values based on the local laboratory reference ranges. Reference ranges provided were global laboratory reference ranges used across all sites. |
| QS | Abbreviation | QS_F01 | | CFQ-R = Cystic fibrosis questionnaire-revised |
| PE | Schedule | PE_L01 | Note: | Either a comprehensive physical examination or a limited physical examination was performed. The limited physical examination included a review of respiratory and cardiovascular body systems at a minimum. |
| RE | Abbreviation | RE_L01 | [1] | FEF2575 = FORCED EXPIRATORY FLOW 25-75% (L); FET = FORCED EXPIRATORY TIME (s); FEV1 = FORCED EXPIRATORY VOLUME IN 1 SECOND (L); FEV1FVC = FEV1/FVC (%); FEV1PP = PERCENT PREDICTED FEV1 (%); FVC = FORCED VITAL CAPACITY (L); FVCPP = PERCENT PREDICTED FVC (%); PEF = PEAK EXPIRATORY FLOW (L); TPEF = TIME TO PEAK EXPIRATORY FLOW (m); VEXT = EXTRAPOLATED VOLUME (m); VEXT/FVC = RATIO OF FEV1 TO FVC (%). |
| RE | Derivation | RE_L02 | Note: | The baseline value was defined as the average of the results from testing on Day $-1$ and at pre-dose on Day 1. |
| RE | Derivation | RE_L03 | Note: | The reference result was the predicted normal result based on age, gender, and height at screening. |
| CM | Dictionary | CM_L01 | Note: | Anatomic Class, Therapeutic Class, and Preferred Name were based on the WHO Drug Global (2020-SEP) coding dictionary. |
| CM | Definition | CM_L02 | Note: | Concomitant medications included all medications in use at date of first study drug dose or started after date of first study drug dose, any medications that started prior to the day of first dose of study drug with missing stop date or that were classified as ongoing. Prior medications included all medications that stopped prior to the day of first dose of the study drug or medications that started prior to the day of first dose of study drug with missing stop date. Medications with missing start and stop dates were classified as both prior and concomitant. |

# Translate Bio, Inc. PROTOCOL NUMBER MRT5005-101

## Figure Specifications

VERSION DATE: 26 October 2021

SPONSOR: Translate Bio, Inc. 29 Hartwell Avenue Lexington, MA 02421 Telephone: (617) 945-7361

PREPARED BY: Rho, Inc. 2635 E NC Hwy 54 Durham, NC 27713 Telephone: (919) 408-8000 Fax: (919) 408-0999

## Figure Specifications

#### Table of Contents

| Gener | al Programming Notes |
|---|---|
| F | igure 14.3.9.1.2 (RE FAH F X) Percent Predicted FEV1 Values by Dose Group, Subject, and Visit |
| F | igure 14.3.9.2.2 (RE FAI F A) Percent Predicted FEV1 Values to Day 29 by Dose Group, Subject, and Visit |
| F | igure 14.3.9.2.2 (RE FAI F B) Percent Predicted FEV1 Values to Day 57 by Dose Group, Subject, and Visit |
| F | igure 14.3.9.2.2 (RE FAI F D) Percent Predicted FEV1 Values to Day 32 by Dose Group, Subject, and Visit |
| F | igure 14.3.9.3 (RE FAC F X) Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit |
| F | igure 14.3.9.3.1 (RE_FAS_F_A) Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 29 ( |
| | igure 14.3.9.3.1 (RE_FAS_F_B) Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 57 ( |
| F | igure 14.3.9.3.1 (RE_FAS_F_D) Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 32 ( |
| F | igure 14.3.9.4 (RE_FAL_F_X) Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit |
| F. | igure 14.3.9.4.1 (RE_FAM_F_A) Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit to Day 29 |
| F. | igure 14.3.9.4.1 (RE_FAM_F_B) Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit to Day 57 |
| F. | igure 14.3.9.4.1 (RE_FAM_F_D) Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit to Day 32 |
| F | igure 14.3.9.4.2 (RE_FAN_F_X) Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit |
| F. | igure 14.3.9.4.3 (RE_FAP_F_A) Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose |
| | Group and Visit to Day 29 8 |
| F'. | igure 14.3.9.4.3 (RE_FAP_F_B) Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose |
| _ | Group and Visit to Day 57 |
| F'. | igure 14.3.9.4.3 (RE_FAP_F_D) Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose |
| _ | Group and Visit to Day 32 |
| | igure 14.3.4.1.1 (LB_FAA_F_X) C Reactive Protein (mg/L) by Dose Group, Subject, and Visit |
| | igure 14.3.4.1.1.1 (LB_FAJ_F_A) C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 29 |
| | igure 14.3.4.1.1.1 (LB_FAJ_F_B) C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 57 |
| | igure 14.3.4.1.1.1 (LB_FAJ_F_D) C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 32 |
| | igure 14.3.4.2.1 (LB_FAB_F_X) White Blood Cells (x10^9/L) by Dose Group, Subject, and Visit |
| | igure 14.3.4.3.1 (LB_FAC_F_X) Neutrophils/Leukocytes (%) by Dose Group, Subject, and Visit |
| | igure 14.3.5.1.1 (VS_FAA_F_A) Body Temperature Values by Dose Group, Subject, and Visit Through Day / |
| | igure 14.3.5.1.1 (VS_FAA_F_B) Body Temperature Values by Dose Group, Subject, and Visit Through Day 36 |
| F. | Analysis Set |
| | MHQIYƏLƏ UCC |

#### General Programming Notes

The following instructions apply to all figure displays.

#### DISPLAY OUTPUTS FOR EACH PART

Each figure will be produced for each study part (A, B, D) unless otherwise specified. Figures will not be produced for the study overall. Each version of the figure will include the relevant study part in the header and in the figure identifier. For example, LB\_FAA\_F\_X will be identified as LB\_FAA\_F\_A for Part A and will include a header to show 'Part A'. A, B or D will be added to each display number.

#### PROGRAMMER NOTES

Programmer notes appear at the bottom of each figure display shell where applicable.

Dose groups for each part are as follow:

- Part A: MRT5005 8mg, MRT5005 16mg, MRT5005 20mg, MRT5005 24mg, Pooled Placebo
- Part B: MRT5005 8mg, MRT5005 12mg, MRT5005 16mg, MRT5005 20mg, Pooled Placebo
- Part D: MRT5005 4mg, Placebo

#### PAGE FORMATTING

The specifications for the format of each page are page size=47, line size=134, font=Courier, font size=8, and margin = 1.5" top, 1" bottom, left, and right.

"Table Source: <Table Number>" will be printed on the right side of the footer for each figure.

#### PRECISION

No preliminary rounding should be performed; rounding should only occur after analysis. To round, consider digit to right of last significant digit: if < 5 then round down, if  $\ge$  5 then round up. Means, medians, 25th percentiles, 75<sup>th</sup> percentiles, and confidence intervals will be presented with one more decimal place than the precision of the data. Standard deviations will be presented with two more decimal places than the precision of the data. Percentages will be presented with one decimal place. Minimums and maximums will be presented with the same precision as the original data, with a maximum of 4 decimal places.

## Figure 14.3.9.1.2 (RE\_FAH\_F\_X) Percent Predicted FEV1 Values by Dose Group, Subject, and Visit Population: Safety Analysis Set

Part: x
Dose Group: xxx



Note: RE F01

X-axis: Assessment Time

Y-axis: Percent Predicted FEV1

Table Source: RE TAA F X

- 1) Line plot of individual subject percent predicted FEV1 values over time
- 2) Separate page/plot for each part and dose group (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 3) Include screening, baseline and all post-baseline visits
- 4) Include a legend to show subject ID (The placebo subject will be labeled in the legend)
- 5) Y-axis will range from 40%-110%

6) For RE\_FAH\_F\_D, replace footnote RE\_F01 with RE\_F01D

Non-unique figures for RE FAH F X:

Figure 14.3.9.2.2 (RE FAI F A) Percent Predicted FEV1 Values to Day 29 by Dose Group, Subject, and Visit

Population: Safety Analysis Set

Table Source: RE TAA F A

#### Notes:

- 1) Repeat RE FAH with the x-axis subset on visits on or before Day 29 for each Part A dose group: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo.
- 2) Time will be represented proportionally on the x-axis

Figure 14.3.9.2.2 (RE FAI F B) Percent Predicted FEV1 Values to Day 57 by Dose Group, Subject, and Visit Population: Safety Analysis Set

Table Source: RE TAA F B

#### Notes:

- 1) Repeat RE FAH with the x-axis subset on visits on or before Day 57 for each Part B dose group: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo.
- 2) Annotate x-axis to indicate the 5 dosing days using a symbol

Figure 14.3.9.2.2 (RE FAI F D) Percent Predicted FEV1 Values to Day 32 by Dose Group, Subject, and Visit Population: Safety Analysis Set

Table Source: RE TAA F D

#### Notes:

- 1) Repeat RE FAH with the x-axis subset on visits on or before Day 32 for each Part D dose group: 4 mg, Placebo.
- 2) Time will be represented proportionally on the x-axis
- 3) Replace footnote RE F01 with RE F01D
- 4) Time will be represented proportionally on the x-axis.

Figure 14.3.9.3 (RE FAC F X)

Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Population: Safety Analysis Set

Note: RE F01

Table Source: RE TAA F X

- 1) Repeat RE\_FAH for the mean values (including standard error bars) for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo).
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) For RE FAC F D, replace footnote RE F01 with RE F01D

Figure 14.3.9.3.1 (RE FAS F A)

Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 29

Population: Safety Analysis Set

Note: RE F01

Table Source: RE TAA F A

#### Notes:

- 1) Repeat RE\_FAH for the mean values (including standard error bars) with the x-axis subset on visits on or before Day 29 for each Part A dose group: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo.
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Time will be represented proportionally on the x-axis

Figure 14.3.9.3.1 (RE FAS F B)

Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 57

Population: Safety Analysis Set

Note: RE F01

Table Source: RE TAA F B

#### Notes:

- 1) Repeat RE\_FAH for the mean values (including standard error bars) with the x-axis subset on visits on or before Day 57 for each Part B dose group: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo.
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed

Figure 14.3.9.3.1 (RE FAS F D)

Mean and Standard Error of Percent Predicted FEV1 Values by Dose Group and Visit Through Day 32

Population: Safety Analysis Set

Note: RE F01D

Table Source: RE TAA F D

#### Notes:

- 1) Repeat RE\_FAH for the mean values (including standard error bars) with the x-axis subset on visits on or before Day 32 for each dose group: (Part D: 4 mg and Placebo).
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Time will be represented proportionally on the x-axis

Figure 14.3.9.4 (RE FAL F X)

Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit

Population: Safety Analysis Set

Note: RE F01

Table Source: RE\_TAA\_F\_X

X-axis: Assessment Time

Y-axis: Absolute Change from Baseline in ppFEV1

#### Notes:

- 1) Repeat RE\_FAH for mean absolute change from baseline values (including standard error bars) for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1
- 4) Time will be represented proportionally on the x-axis for RE FAL F A and RE FAL F D
- 5) For RE FAH F D, replace footnote RE F01 with RE F01D

Figure 14.3.9.4.1 (RE FAM F A)

Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 29

Population: Safety Analysis Set

Note: RE F01

Table Source: RE\_TAA\_F\_A

X-axis: Assessment Time

Y-axis: Absolute Change from Baseline in ppFEV1

#### Notes:

- 1) Repeat RE\_FAH for mean absolute change from baseline values (including standard error bars) for each dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, and Pooled Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1 up to Day 29
- 4) Time will be represented proportionally on the x-axis

Figure 14.3.9.4.1 (RE FAM F B)

Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 57

Population: Safety Analysis Set

Note: RE F01

Table Source: RE\_TAA\_F\_B

X-axis: Assessment Time

Y-axis: Absolute Change from Baseline in ppFEV1

- Repeat RE\_FAH for mean absolute change from baseline values (including standard error bars) for each dose group: (Part: 8 mg, 12 mg, 16 mg, 20 mg and Pooled Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1 up to Day 57

Figure 14.3.9.4.1 (RE FAM F D)

Mean and Standard Error of Absolute Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 32

Population: Safety Analysis Set

Note: RE F01D

Table Source: RE\_TAA\_F\_D

X-axis: Assessment Time

Y-axis: Absolute Change from Baseline in ppFEV1

#### Notes:

- 1) Repeat RE\_FAH for mean absolute change from baseline values (including standard error bars) for each dose group: (Part D: 4 mg and Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1 up to Day 32
- 4) Time will be represented proportionally on the x-axis

Figure 14.3.9.4.2 (RE FAN F X)

Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit
Population: Safety Analysis Set

Note: RE F01

Table Source: RE TAB F X

X-axis: Assessment Time

Y-axis: Relative Change from Baseline in ppFEV1 (%)

#### Notes:

- 1) Repeat RE\_FAH for mean relative change from baseline values (including standard error bars) for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 20 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1.
- 4) Time will be represented proportionally on the x-axis for RE FAN F A and RE FAN F D.
- 5) For RE FAN F D, replace footnote RE F01 with RE F01D

Figure 14.3.9.4.3 (RE FAP F A)

Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 29

Population: Safety Analysis Set

Note: RE F01

Table Source: RE\_TAB\_F\_A

X-axis: Assessment Time

Y-axis: Relative Change from Baseline in ppFEV1 (%)

#### Notes:

- 1) Repeat RE\_FAH for mean relative change from baseline values (including standard error bars) for each dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, and Pooled Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1 up to Day 29.
- 4) Time will be represented proportionally on the x-axis

Figure 14.3.9.4.3 (RE\_FAP\_F\_B)

Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 57
Population: Safety Analysis Set

Note: RE F01

Table Source: RE\_TAB\_F\_B

X-axis: Assessment Time

Y-axis: Relative Change from Baseline in ppFEV1 (%)

#### Notes:

- Repeat RE\_FAH for mean relative change from baseline values (including standard error bars) for each dose group: (Part B: 8 mg, 12 mg, 16 mg, 20 mg and Pooled Placebo)
- 2) Plot is only created for Part B
- 3) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 4) Include all visits after the pre-dose measure on Day 1 up to Day 57.

Figure 14.3.9.4.3 (RE\_FAP\_F\_D)

Mean and Standard Error of Relative Change from Baseline in Percent Predicted FEV1 Values by Dose Group and Visit to Day 32

Population: Safety Analysis Set

Note: RE F01D

Table Source: RE TAB F D

X-axis: Assessment Time

Y-axis: Relative Change from Baseline in ppFEV1 (%)

- 1) Repeat RE\_FAH for mean relative change from baseline values (including standard error bars) for each dose group: (Part D: 4 mg and Placebo)
- 2) Note that all values will display on the same plot and the 'Dose Group' header will be removed
- 3) Include all visits after the pre-dose measure on Day 1 to Day 32.
- 4) Time will be represented proportionally on the x-axis

Figure 14.3.4.1.1 (LB\_FAA\_F\_X) C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Population: Safety Analysis Set

Table Source: LB TAA F X

X-axis: Assessment Time

Y-axis: C Reactive Protein (mg/L)

#### Notes:

- 1) Line plot of individual subject CRP values over time
- 2) Separate page/plot for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 3) Include screening, baseline and all post-baseline visits
- 4) Y-axis minimum value will be zero, maximum will be 90
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.4.1.1.1 (LB\_FAJ\_F\_A)

C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 29

Population: Safety Analysis Set

Table Source: LB TAA F A

X-axis: Assessment Time

Y-axis: C Reactive Protein (mg/L)

#### Notes:

- 1) Line plot of individual subject CRP values over time
- 2) Separate page/plot for each dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo)
- 3) Include screening, baseline and all post-baseline visits through Day 29
- 4) Y-axis minimum value will be zero, maximum will be 90
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.4.1.1.1 (LB\_FAJ\_F\_B)

C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 57

Population: Safety Analysis Set

Table Source: LB TAA F B

X-axis: Assessment Time

Y-axis: C Reactive Protein (mg/L)

- 1) Line plot of individual subject CRP values over time
- 2) Separate page/plot for each dose group: (Part B: 8 mg, 12 mg, 16 mg, 20 mg and Pooled Placebo)
- 3) Include screening, baseline and all post-baseline visits through Day 57

- 4) Y-axis minimum value will be zero, maximum will be 90
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.4.1.1.1 (LB\_FAJ\_F\_D)

C Reactive Protein (mg/L) by Dose Group, Subject, and Visit Through Day 32

Population: Safety Analysis Set

Table Source: LB TAA F D

X-axis: Assessment Time

Y-axis: C Reactive Protein (mg/L)

#### Notes:

- 1) Line plot of individual subject CRP values over time
- 2) Separate page/plot for each dose group: (Part D: 4 mg and Placebo)
- 3) Include screening, baseline and all post-baseline visits through Day 32
- 4) Y-axis minimum value will be zero, maximum will be 90
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.4.2.1 (LB\_FAB\_F\_X) White Blood Cells (x10^9/L) by Dose Group, Subject, and Visit Population: Safety Analysis Set

Table Source: LB TAB F X

X-axis: Assessment Time

Y-axis: White Blood Cells (x10^9/L)

#### Notes:

- 1) Line plot of individual subject WBC values over time
- 2) Separate page/plot for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 3) Include screening, baseline and all post-baseline visits
- 4) Y-axis range will be 3 to 19
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.4.3.1 (LB\_FAC\_F\_X) Neutrophils/Leukocytes (%) by Dose Group, Subject, and Visit Population: Safety Analysis Set

Table Source: LB\_TAB\_F\_X

X-axis: Assessment Time

Y-axis: Neutrophils/Leukocytes (%)

#### Notes:

- 1) Line plot of individual subject neutrophil values over time
- 2) Separate page/plot for each part and dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, Pooled Placebo; Part B: 8 mg, 12 mg, 16 mg, 20 mg, Pooled Placebo; Part D: 4 mg, Placebo)
- 3) Include screening, baseline and all post-baseline visits
- 4) Y-axis range will be 5% 90%
- 5) Time will be represented proportionally on the x-axis

Figure 14.3.5.1.1 (VS\_FAA\_F\_A)

Body Temperature Values by Dose Group, Subject, and Visit Through Day 7

Population: Safety Analysis Set

Table Source: VS\_TAA\_F\_A

X-axis: Assessment Time
Y-axis: Temperature (C)

#### Notes:

- 1) Line plot of individual subject temperature values over time
- 2) Separate page/plot for each dose group: (Part A: 8 mg, 16 mg, 20 mg, 24 mg, and Pooled Placebo)
- 3) Include baseline and only visits through Day 7 for Part A.
- 4) Y-axis range will be 35(C) 40(C)

Figure 14.3.5.1.1 (VS\_FAA\_F\_B)
Body Temperature Values by Dose Group, Subject, and Visit Through Day 36
Population: Safety Analysis Set

Table Source: VS\_TAA\_F\_B
X-axis: Assessment Time
Y-axis: Temperature (C)

#### Notes:

- 1) Line plot of individual subject temperature values over time
- 2) Separate page/plot for each dose group: (Part B: 8 mg, 12 mg, 16 mg, 20 mg and Pooled Placebo)
- 3) Include baseline and only visits through Day 36 for Part B.
- 4) Y-axis range will be 35(C) 40(C)

Figure 14.3.5.1.1 (VS\_FAA\_F\_D)

Body Temperature Values by Dose Group, Subject, and Visit Through Day 11

Population: Safety Analysis Set

X-axis: Assessment Time Y-axis: Temperature (C)

Table Source: VS TAA F D

- 1) Line plot of individual subject temperature values over time
- 2) Separate page/plot for each dose group: (Part D: 4 mg and Placebo)
- 3) Include baseline and only visits through Day 11 for Part D.
- 4) Y-axis range will be 35(C) 40(C)

#### Footnotes

| Data | Footnote | | | |
|---|---|---|---|---|
| Type | Type | Code | Prefix | Footnote |
| RE | Baseline | RE F01 | Note: | The baseline value was defined as the average of the results from testing on Day -1 |
| | | _ | | and at pre-dose on Day 1. |
| RE | Baseline | RE F01D | [1] | The baseline value was defined as the result from testing pre-dose on Day 1. |

### **Certificate Of Completion**

Envelope Id: B73E49A7E969424D8251CBFC3DA6A5E8

Subject: Please DocuSign: MRT5005-101\_CSR\_SAP\_v1.0\_26OCT2021.pdf

Source Envelope:

Document Pages: 49 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

**Envelope Originator:** 



### **Record Tracking**

Status: Original

10/26/2021 12:35:33 PM

Security Appliance Status: Connected Storage Appliance Status: Connected Holder:

Signatures: 3

Initials: 0

Pool: FedRamp

Pool: Rho, Inc.

Location: DocuSign

Location: DocuSign

## **Signer Events**

### Signature

## **Timestamp**

Sent: 10/26/2021 12:37:12 PM Viewed: 10/26/2021 2:15:25 PM Signed: 10/26/2021 2:16:16 PM

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

2302C1A3-4255-4335-B26A-9E3BCC08FC15

Using IP Address: 108.49.127.187

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

### **Electronic Record and Signature Disclosure:**

Accepted: 10/30/2020 6:29:38 PM

ID: 9dc2171d-a1a9-4bcb-981c-5e73974e4d39

Sent: 10/26/2021 12:37:12 PM Viewed: 10/26/2021 4:01:29 PM Signed: 10/26/2021 4:02:34 PM

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

ECE62283-4997-4BFA-AB04-AFB2B0B4805A

Using IP Address: 24.62.27.123

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 4/28/2020 12:50:56 PM

ID: 779ae970-3904-4e59-8f54-e10a5db28185

Signer Events Signature

**Timestamp**Sent: 10/26/2021 12:37:11 PM
Viewed: 10/26/2021 12:37:34 PM
Signed: 10/26/2021 12:38:06 PM

Rho, Inc.

Security Level: Email, Account Authentication (Required)

Signature Adoption: Pre-selected Style

Signature ID:

E8BC91C1-B54B-4472-9F4A-53C7CA804C98

Using IP Address: 4.34.23.236

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

## **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

| In Person Signer Events | Signature | Timestamp |
|---|---|---|
| Editor Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Witness Events | Signature | Timestamp |
| Witness Events Notary Events | Signature Signature | Timestamp |
| | _ | · |
| Notary Events | Signature | Timestamp |
| Notary Events Envelope Summary Events Envelope Sent Certified Delivered Signing Complete | Signature Status Hashed/Encrypted Security Checked Security Checked | Timestamps 10/26/2021 12:37:12 PM 10/26/2021 12:37:34 PM 10/26/2021 12:38:06 PM |

### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Rho, Inc. (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

## Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

## Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### How to contact Rho, Inc.:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: rho-css@rhoworld.com

## To advise Rho, Inc. of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at rho-css@rhoworld.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

### To request paper copies from Rho, Inc.

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to rho-css@rhoworld.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

## To withdraw your consent with Rho, Inc.

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to rho-css@rhoworld.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

## Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Rho, Inc. as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Rho, Inc. during the course of your relationship with Rho, Inc..